## STATISTICAL ANALYSIS PLAN

An open-label, multi-center, follow-up trial to evaluate the long-term safety and efficacy of privaracetam (ucb 34714) used as adjunctive treatment at a flexible dose up to a maximum of 200mg/day in subjects aged 16 years or older suffering from epilepsy

**SAP/Amendment Number** 

Final SAP

SAP Amendment 1

27 January 2014

11 February 2019

### **Confidentiality Material**

### Confidential

This document is the property of UCB and may not – in full or in part – be passed on, reproduced, published, or otherwise used without the express permission of UCB. This document

# **TABLE OF CONTENTS**

| LI | ST OF ABB | REVIATIONS | 6 |
|---|---|---|---|
| 1 | INTRODU | UCTION | 8 |
| 2 | PROTOC | OL SUMMARY | 8 |
| | 2.1 Stud | dy objectives | 8 |
| | 2.1.1 | Primary objective | 8 |
| | 2.1.2 | Secondary objectives | 8 |
| | 2.1.3 | Exploratory objectives | ;011 |
| | 2.2 Stud | OL SUMMARY dy objectives Primary objective Secondary objectives Exploratory objectives dy variables Safety variables 1.1 Primary safety variables 1.2 Other safety variables Efficacy variables 2.1 Secondary efficacy variables Pharmacoeconomic variables Pharmacoeconomic variables dy Design and Conduct ermination of Sample Size NALYSIS CONSIDERATIONS heral presentation of summaries and analyses | 8 |
| | 2.2.1 | Safety variables | 8 |
| | 2.2. | 1.1 Primary safety variables | 8 |
| | 2.2. | 1.2 Other safety variables | 9 |
| | 2.2.2 | Efficacy variables | 9 |
| | 2.2. | 2.1 Secondary efficacy variables | 9 |
| | 2.2. | 2.2 Other efficacy variables | 9 |
| | 2.2.3 | Pharmacoeconomic variables Constant Con | 10 |
| | 2.3 Stud | dy Design and Conduct | 10 |
| | 2.4 Det | ermination of Sample Size | 14 |
| 3 | DATA Al | NALYSIS CONSIDERATIONS | 14 |
| | 3.1 Gen | neral presentation of summaries and analyses | 14 |
| | 3.2 Ana | alysis time points | |
| | 3.2.1 | First and last dose of BRV | 14 |
| | 3.2.2 | Relative day | 14 |
| | 3.2.3 | Summaries at Study Entry | 15 |
| | 3.2.4 | Study periods | 16 |
| | 3.2.5 | Monthly time intervals | |
| | ~ | Last Value on BRV Treatment | 17 |
| | 3.20 | Exposure duration and exposure duration cohorts | 18 |
| | 3.2.8<br>3.3 Def | Study visit cohorts | 18 |
| , | 3.3 Def | inition of Baseline Values | 18 |
| er | 3.4 Pro | tocol deviations | 18 |
| | 3.5 Ana | alysis Sets | 19 |
| | 3.5.1 | Safety Analysis Set | 19 |
| | 3.5.2 | Efficacy Analysis Sets | 19 |
| | 3.6 Trea | atment Assignment and Treatment Groups | 19 |

| UCB<br>Statistical Analysis | s Plan Brivaracetam | 11 February 2019<br>N01125 |
|---|---|---|
| • | | |
| 6.4.3 | History of previous AED use | |
| 6.4.4 | AEDs taken at study entry | 29 |
| | EMENTS OF TREATMENT COMPLIANCE | 29 |
| | Y ANALYSES | 29 |
| | istical analyses of secondary efficacy variables | 29 |
| 8.1.1 | EMENTS OF TREATMENT COMPLIANCE Y ANALYSES | 30 |
| 8.1.2 | Percent reduction in POS frequency | 30 |
| 8.1.3 | Responder outcome for POS frequency | 30 |
| 8.2 Ana | lysis of other efficacy variables | 30 |
| 8.2.1 | Subjects with partial onset seizures | 30 |
| 8.2.1 | 1.1 Specified Month seizure freedom | 31 |
| 8.2.2 | Subjects with Primary Generalized Seizures | 31 |
| 8.2.2 | 2.1 All type seizure days | 31 |
| 8.2.2 | Percent reduction in all type seizure days | 31 |
| 8.2.2 | 2.3 Responder outcome for all type seizure days | 31 |
| 8.2.2 | 2.4 Specified month seizure freedom | 31 |
| 8.2.3 | QOLIE-31-P | 32 |
| 8.2.4 | 2.4 Specified month seizure freedom | 32 |
| 8.2.5 | Direct cost parameters | 33 |
| 8.2.6 | Indirect cost parameters | 33 |
| 8.2.7 | The number of school of working days lost will not be sumn | narized but |
| | will be provided in subject data listings. Socio-professional | |
| | COKINETICS AND PHARMACODYNAMICS | |
| 10 IMMUNO | LOGICAL PROCEDURES | 34 |
| 11 SAFETY | ANALYSES. | |
| II.I EXIC | ent of exposure | |
| | erse events | |
| / | Definition of treatment-emergent AE | |
| 11.2.2 | | |
| 11.3 Clin | ical laboratory evaluations | 36 |
| 11.3 Clin<br>11.3.1<br>11.3.2<br>11.3.3 | Hematology and blood chemistry parameters | 37 |
| 11.3.2 | Macroscopic urinalysis | 37 |
| 11.3.3 | Microscopic urinalysis | 38 |
| 11.4 Vita | l signs, physical findings, and other observations related to saf | ety38 |
| 11.4.1 | Vital signs | 38 |
| 11.4.2 | Electrocardiograms | 39 |

| UCB<br>Statistical Analysis | Plan Brivaracetam | 11 February 2019<br>N01125 |
|---|---|---|
| 11.4.3 | Physical examination | 39 |
| 11.4.4 | Neurological examination | |
| 11.4.6 | HADS | 39 |
| 11.4.7 | Columbia-Suicide Severity Rating Scale | 40 Single |
| 12 REFERENCE | CES | 41 iOns |
| 13 APPENDIC | ES | 43i <sup>(2)</sup> |
| 13.1 OOL | Psychiatric and mental status HADS Columbia-Suicide Severity Rating Scale ES E-31-P total and subscale score calculations ct site transfers Criteria Hematology parameters | 42 |
| 13.1 QOD | ct site transfers | ~ 44 |
| 13.2 Buoje | criteria | 25 45 |
| 13.3 1 | Hematology parameters | 45 |
| 13.3.1 | Blood chemistry parameters | 46 |
| 13.3.2 | Urinalysis | 48 |
| 13.3.3 | Vital signs and hody weight | 48 |
| This document cannot be use | Columbia-Suicide Severity Rating Scale ES ES E-31-P total and subscale score calculations ct site transfers criteria | |

### LIST OF ABBREVIATIONS

AΕ adverse event **AED** antiepileptic drug antimyoclonic drug **AMD ALP** Alkaline phosphatase **ALT** alanine aminotransferase aspartate aminotransferase AST **ATC Anatomic Therapeutic Class** 

BMI body mass index bpm Beats per minute **BRV** brivaracetam **BUN** blood urea nitrogen

iensions or variations thereof. Committee for Medicinal Products for Human Use **CHMP** 

CR CL creatinine clearance **CRF** case report form

Columbia-Suicide Severity Rating Scale C-SSRS

**DBP** diastolic blood pressure electrocardiogram **ECG** Early Discontinuation Visit **EDV** EQ-5D EuroQol 5 Dimensions ER emergency room

European Union EU F Female

Food and Drug Administration **FDA** 

**FEV** Full Evaluation Visit

Final Visit FV

**GGT** Gamma-glutamyl transpeptidase Hospital Anxiety and Depression Scale **HADS** 

HDL High-density lipoprotein Health-Related Quality of Life **HROoL** 

**ILAE** International League Against Epilepsy

low-density lipoprotein LDL

MedDRA Medical Dictionary for Regulatory Activities

M Male

MEV Minimal Evaluation Visit

Not applicable placebo

potentially clinically significant treatment-emergent

primary generalized seizures

PBO PGS PGS partial onset seizure preferred term

Patient Weighted Quality of Life in Epilepsy OOLIE-31-P

Questionnaire

11 February 2019 **UCB** N01125 Statistical Analysis Plan Brivaracetam Red Blood Cell **RBC SAE** serious adverse event **SAP SBP** SD **SEV SGOT SGPT** SOC **TEAE** ULD ULN anization Drug on Visit on Visit on Visit and Recapiled authorization applied to support any marketing authorization applied to support any marketing authorization applied to support any marketing authorization and the use of the support any marketing authorization. V VAS

#### 1 INTRODUCTION

This statistical analysis plan (SAP) defines the scope of statistical analyses and provides a or variations thereof detailed description of statistical methodology for the statistical analyses to support the final clinical study report for N01125.

#### 2 PROTOCOL SUMMARY

#### 2.1 Study objectives

#### 2.1.1 **Primary objective**

To evaluate the long-term safety and tolerability of brivaracetam (BRV) at individualized doses with a maximum of 200mg/day in subjects suffering from epilepsy

#### 2.1.2 Secondary objectives

To evaluate the maintenance of efficacy over time of BRV (for subjects with partial onset seizures [POS] and subjects with primary generalized seizures [PGS])

No secondary efficacy objectives are defined for subjects with Unverricht-Lundborg Disease (ULD) or subjects entering the study from N01315.

### 2.1.3 **Exploratory objectives**

Exploratory objectives for subjects with POS/PGS

- To explore direct medical resource use and indirect cost parameters for the first 2 years
- To obtain a description of the subject's self-reported health status for the first 2 years
- To explore the effects of BRV on the subject's Health-Related Quality of Life (HRQoL), anxiety, and depression for the first 2 years
- To explore any change in the subject's socio-professional status for the first 2 years

No exploratory objectives are defined for ULD subjects or subjects entering the study from 01315.

### Study variables 2.2

#### 2.2.1 Safety variables

Note: Assessments specified as performed within the first 2 years of the Evaluation Period are not applicable to subjects entering the study from N01315.

### 2.2.1.1 Primary safety variables

- Occurrence of a treatment-emergent adverse event (TEAE)
- Withdrawal due to adverse event (AE)
- Occurrence of a serious adverse event (SAE)

#### 2.2.1.2 Other safety variables

- Laboratory tests (hematology, blood chemistry, urinalysis)

- Inysical and neurological examinations

  Change in Hospital Anxiety and Depression Scale (HADS) scores from the Baseline of the previous study to each assessment for the first 2 years and to the last Evaluation Period assessment during the first 2 years

  Efficacy variables

  2.2.2 Efficacy variables

  2.2.2.1 Second

For subjects with focal-onset epilepsy:

- POS (type I) frequency per 28 days during the Evaluation Period
- Percent reduction in POS (type I) frequency per 28 days from Baseline of the previous study to the Evaluation Period
- Responder rate for POS (type I) frequency over the Evaluation Period. A responder is defined as a subject with a  $\geq$ 50% reduction in seizure frequency from the Baseline Period of the previous study.

No secondary efficacy variables are defined for subjects with generalized epilepsy or subjects with ULD or subjects entering the study from N01315.

### 2.2.2.2 Other efficacy variables

For subjects with focal-onset epilepsy:

Percentage of subjects continuously seizure-free for all seizure types (I+II+III) for at least 6 months and at least 12 months during the Evaluation Period

For subjects with generalized epilepsy:

- Generalized (type II) seizure days per 28 days during the Evaluation Period
- Percent reduction in generalized (type II) seizure days per 28 days from Baseline of the previous study to the Evaluation Period
- Responder rate for generalized (type II) seizure days over the Evaluation Period. A responder is defined as a subject with a  $\geq$ 50% reduction in seizure days from the Baseline Period of the previous study.
- Percentage of subjects continuously seizure-free for all seizure types (I+II+III) for at least 6 months and at least 12 months during the Evaluation Period

The following will be evaluated separately for subjects with focal-onset epilepsy and subjects with generalized epilepsy:

- EuroQol 5 Dimensions (EQ-5D) questionnaire response for each assessment for the first 2 years 2 years for the Evaluation Period and for the last assessment during the first 2 years Evaluation Period Change in Patient Weighted Quality of Life in Epilepsy Questionnaire (QOLIE-31-P)

#### 2.2.3 Pharmacoeconomic variables

Due to the inconsistencies in data captured and collection forms across LTFU studies, the following variables will be provided in subject data listings only, but will not be evaluated or descriptive summarized:

- Direct costs (healthcare provider consultations not foreseen by the protocol, concurrent medical procedures, concomitant medications, hospitalizations, and emergency room [ER] visits) during the first 2 years of the Evaluation Period
- Indirect costs (work days or school days lost by the subject and days subject received help from a caregiver) during the first 2 years of the Evaluation Period
- Socio-professional data for each assessment for the first 2 years and for the last assessment during the first 2 years of the Evaluation Period

No pharmacoeconomic variables are defined for ULD subjects or subjects entering the study from N01315.

# Study Design and Conduct 2.3

This is an open-label, long-term follow-up, multicenter, noncomparative, single-arm study of BRV. The primary objective is to evaluate the long-term safety and tolerability of BRV at individualized doses up to a maximum of 200mg/day in subjects with epilepsy. The secondary objective is to evaluate the maintenance of efficacy of BRV. Exploratory objectives are to assess the effects of BRV on subjects' HRQoL, obtain information on the direct and indirect costs, and explore changes in socio-professional status.

N01125 enrolled subjects 16 years of age and older who had completed N01114, N01252 (non-Indian subjects only), N01254 (non-Indian subjects only), N01187, or N01236. N01114 and N01252 enrolled subjects with focal-onset seizures with or without secondary generalization (designated as "POS subjects"). N01254 enrolled subjects with focal-onset epilepsy and a smaller number of subjects with generalized epilepsy (designated as "PGS subjects"). N01187 and N01236 enrolled subjects with ULD. Subjects entering the study from long-term follow-up study (N01315) were 16 years of age and older with from POS.

Subjects from double-blind, placebo-controlled studies N01114, N01187, and N01236 were to enter N01125 at a dose of 100mg/day after completion of a blinded Conversion Period. Subjects from double-blind, placebo-controlled N01252 were to enter N01125 at a dose of

50mg/day. The starting doses for subjects from double-blind, placebo-controlled, flexibledose study N01254 were based on the blinded dose levels achieved during the Maintenance Period of N01254 but were not to exceed 100mg/day; thus, starting doses for subjects from

Subjects who enrolled in the study entered an Evaluation Period during which treatment with BRV was initiated. The dose of BRV can be adjusted based on the individual subject's seizure control and tolerability. Dose increases can be made in increments of 50mg/day on a weekly basis up to a maximum of 200mg/day: dose doors 50mg/day on a weekly basis up to a maximum of 200mg/day: dose doors to be made in increments of 50mg/day on a weekly basis up to a maximum of 200mg/day: dose doors to be made in increments of 50mg/day on a weekly basis up to a maximum of 200mg/day; dose doors to be made in increments of 50mg/day on a weekly basis up to a maximum of 200mg/day; dose doors to be made in increments of 50mg/day on a weekly basis up to a maximum of 200mg/day; dose doors to be made in increments of 50mg/day on a weekly basis up to a maximum of 200mg/day; dose doors to be made in increments of 50mg/day on a weekly basis up to a maximum of 200mg/day; dose doors to be made in increments of 50mg/day on a weekly basis up to a maximum of 200mg/day; dose doors to be made in increments of 50mg/day on a weekly basis up to a maximum of 200mg/day; dose doors to be made in increments of 50mg/day on a weekly basis up to a maximum of 200mg/day; dose doors to be made in increments of 50mg/day on a weekly basis up to a maximum of 200mg/day; dose doors to be made in increments of 50mg/day on a weekly basis up to a maximum of 200mg/day on a weekly basis up to a weekly basis up to a 50mg/day on a weekly basis. Subjects who discontinue treatment with BRV enter a Down-Titration Period during which the dose of BRV is decreased in steps of 50mg/day with a last down-titration step at 20mg/day for 1 week. Subjects who have completed the Down-Titration Period or subjects who discontinue during the Evaluation Period without entering the Down-Titration Period enter a Post-Treatment Period for a minimum of 2 weeks and a maximum of 4 weeks.

The maximum allowable daily dose for this study was increased from 150mg/day to 200mg/day based on integrated amendment 25 to the protocol It is recommended that the daily dose be administered in 2 equal intakes.

Dose adjustment to concomitant antiepileptic drugs (AEDs) may be made at any time during the study and subjects may start new AEDs. Concomitant AEDs may also be discontinued; however, special considerations apply if the discontinuation of such AEDs results in the subject receiving BRV monotherapy. Previously, in the event of excellent efficacy and tolerability of BRV, withdrawal of concomitant AEDs resulting in monotherapy of BRV may have been attempted by the Investigator for subjects with POS or PGS. With integrated amendment 25 to the protocol, conversion to monotherapy is no longer permitted; however, subjects already on BRV monotherapy are allowed to continue monotherapy treatment. No conversion to monotherapy is permitted for subjects with ULD.

The visit schedule for this study depends on the previous study from which the subject was enrolled and the numbering of study visits differs depending on the previous study. Study visits at Months 6, 12518, 24, and so forth are either Full Evaluation Visits (FEVs) or Yearly Evaluation Visits (YEVs) at which a greater number of assessments are performed for all subjects from previous studies. For subjects coming from N01114, study visits at Months 1, 3, 5, 15, 21 are Minimal Evaluation Visits (MEVs) at which few assessments are generally performed. Study visits at Months 2, 4, and 9 are FEVs. For subjects coming from N01252, N01254, N01187, and N01236, study visits at Months 1, 3, 9, 15, and 21 are MEVs. The study visit at Month 2 is an FEV. In addition, a phone call is scheduled at the end of the Down-Titration Period and a Drug-Free Final Visit (FV) is scheduled at the end of the Post-Treatment Period. The study schedule, as just described, is shown in Table 2–1 and Table 2–

Table 2–1: Study Schedule for Subjects from N01114, N01252, and N01254

| Subjects coming from Exploratory Studies (N01114) | | | | ing from Conf<br>(N01252, N012 | irmatory Studies<br>254) |
|---|---|---|---|---|---|
| Month | Visit | Type of Visit | Month | Visit | Type of Visit |
| | 1st year Follov | v-up | - | l <sup>st</sup> year Follow | -up |
| МО | V1 | Entry Visit | МО | V1 | Entry Visit |
| M1 | V2 | MEV | M1 | V2 | MEV |
| M2 | V3 | FEV | M2 | V3 | FEV |
| M3 | V4 | MEV | M3 | V4 | MEV |
| M4 | V5 | FEV | M4 | -9 SU3 | |
| M5 | V6 | MEV | M5 | " sugar | |
| M6 | V7 | FEV | M6 | dil <sup>O</sup> V5 | FEV |
| M7 | | | -M7 opli | | |
| M8 | | | M8 | | |
| M9 | V8 | FEV | √2 M9 | V6 | MEV |
| M10 | | EDP SUR | M10 | | |
| M11 | | DEL DO DE | M11 | | |
| 2nd and subsequent years Follow-up | | | 2nd and su | ıbsequent yea | rs Follow-up |
| M12 | V9 | YEV | M12 | V7 | YEV |
| M15 | V10 | MEV MEV | M15 | V8 | MEV |
| M18 | V11 0 | FEV | M18 | V9 | FEV |
| M21 | V12) | MEV | M21 | V10 | MEV |

FEV=Full Evaluation Visit; MEV=Minimal Evaluation Visit; M=month; V=Visit; YEV=Yearly Evaluation Visit

Study Schedule for Subjects from N01187 and N01236 **Table 2–2:** 

| Subjects coming from ULD Confirmatory Studies (N01187, N01236) | | |
|---|---|---|
| Month | Visit | Type of Visit |
| | 1st year Follow | -up |
| M0 | V1 | Entry Visit |
| M1 | V2 | MEV |
| M2 | V3 | FEV : OTS |
| M3 | V4 | MEV MEV |
| M4 | | 201 |
| M5 | | 92 |
| M6 | V5 | FEV |
| M7 | | · calil |
| M8 | Õ | 4 along |
| M9 | V6 CO. | MEV |
| M10 | V6 | |
| M11 | ORO INFO | |
| | 2 <sup>nd</sup> and subsequent years Follow-up | |
| M12 | JO V7 | YEV |
| M15 | V8 | MEV |
| M18 | V9 | FEV |
| M21 | V10 | MEV |
| SUP | | |

FEV=Full Evaluation Visit; MEV=Minimal Evaluation Visit; M=month; ULD=Unverricht-Lundborg disease; V=Visit; YEV=Yearly Evaluation Visit

All subjects should have a Visit 1 at the start of N01125. Visit 1 will typically correspond to the last visit from the previous study and should be the visit at which study drug is dispensed Entry Visit (SEV) at the time of entry into N01125.

Subjects entering from N01315 will a same time their F. for N01125. However, some subjects had a delay in treatment with study drug after completion of the previous study. Such subjects may have had an additional Supplemental

Subjects entering from N01315 will perform their Last Visit in N01315 and perform at the same time their First Visit in N01125. They will follow the schedule of 1 visit/3months: 1 Full Evaluation Visit alternating with 1 Minimal Evaluation Visit. Yearly Evaluation Visit will be performed in replacement of the first Full Evaluation Visit of each year.

This study will run throughout the duration of the clinical development period of BRV, and In all an increatory POS, whether or not sponsor decides to close the study, until a managed access program, named patient program, compassionate use program, or similar type of access program is established as allowed per country-specific requirement in addition to legal and regulatory guidelines, or until BRV development is stopped by the Sponsor.

2.4 Determination of Sample Size

No sample size will continue until a marketing authorization is granted by any Health Authority in an

No sample size calculation was done. Sample size was dependent upon recruitment into and completion of preceding studies. At the time of development of this SAP amendment 1, the enrollment into this study has been completed; a total of 859 subjects were enrolled into N01125 including 6 subjects entering the study from N01315.

### DATA ANALYSIS CONSIDERATIONS 3

### General presentation of summaries and analyses 3.1

Statistical analysis and generation of tables, figures, subject data listings, and statistical output will be carried out using SAS® Version 9.1 or higher.

Descriptive statistics, such as the mean, standard deviation (SD), median, 25th percentile, 75th percentile, minimum value, and maximum value for quantitative variables, and counts and percentages for categorical variables, will be provided. Denominators for percentages will generally be based on the set of subjects with at least 1 assessment at the time point or at least 1 assessment during the time interval being summarized.

All summaries will be descriptive; no statistical hypothesis testing is planned.

Unless otherwise noted, summaries will present BRV overall, which will include all subjects exposed to BRV during the study.

Subject data listings will be provided and will present source data and key derived variables for statistical analyses.

### **Analysis time points** 3.2

## First and last dose of BRV 3.2.1

Unless otherwise noted, all references to the first dose of BRV in this SAP refer to the first dose of BRV during N01125 (ie, not the first dose of BRV from the previous study in which subjects participated in prior to N01125). Unless otherwise noted, all references to the last known dose of BRV in this SAP refer to the last dose of BRV taken across any study periods (ie, the last dose of BRV across both the Evaluation and Down-Titration Periods).

#### 3.2.2 Relative day

Relative day will be calculated as the current date minus the date of first dose of study drug for days prior to the first dose of study drug, and the current date minus the date of first dose

of study drug plus 1 for days on or after the day first dose of study drug and prior to or on the day of last study drug dose (eg, the day of first dose will be Day 1 and the day prior to first dose will be Day -1), ie, Day 1 representing the day of first dose of BRV, the previous day is and the last dose of BRV, relative days to Day 1

as the current date minus the date of last dose of BRV and including a '+' to denote post treatment days (eg, the day after the last dose of BRV will be Day +1). Relative day will not be calculated for partial or missing dates.

3.2.3 Summaries at Study France.

Study Entry denotes an analysis time point that will summarize assessments done at the last visit of the previous study for most subjects as described below, but may also include assessments that may have been performed at Supplemental Entry Visits (SEVs) for some subjects who did not immediately enter N01125.

There are 4 groups of subjects to consider:

- 1. Subjects who immediately entered N01125 after completing the Treatment Periods for N01252 and N01254 or the blinded Conversion Periods for N01114, N01187, and N01236
- 2. Subjects who entered the Down-Titration Period of the previous study and entered N01125 during the Down-Titration Period
- 3. Subjects who did not immediately enter N01125 and had a gap in treatment with study drug between the previous study and N01125Subjects
- 4. Subjects entering the study from N01315 who entered after their N01315 study sites were closed

Subjects in Categories 1 and 2
Subjects in categories 1 and 2 will generally not have any interruption in study drug dosing during the transition to N01125. For such subjects, selected assessments from the following visits from the previous study will be summarized at Study Entry:

| Visit (Time Point) |
|--------------------|
| Visit 9 (Week 16) |
| Visit 10 (Week 12) |
| Visit 7 (Week 12) |
| Visit 8 (Week 16) |

The following assessments were to be performed for all subjects at the above time points: laboratory parameters, vital signs, and ECGs; these assessments will be summarized at Study Entry. The following assessments were to be performed for all subjects from N01252 and N01254 at the above time points: QOLIE-31-P, HADS, EQ-5D and socio-professional data; however, these assessments will not be summarized at Study Entry.

Subjects in Category 3

Some subjects in category 3 have data available from an SEV at the time of entry into N01125. Laboratory parameters, vital signs, and ECGs collected at SEV will be summarized Brivaracetam

at Study Entry. If one or more of these assessments were not performed at SEV, or if a subject in category 3 does not have an SEV, then the subject will be excluded from summaries of Study Entry for the assessments that were not performed.

Subjects in category 4 will have their demographic data including date of birth, country, gender, race, and ongoing medication data transferred into N01125. Laboratory parameters, vital signs, and ECGs collected at SEV will be collected at Study Entry.

3.2.4 Study periods

The study is divided into 3 periods: Evaluation Period, Down-Titration Period and CDES case report form (CDES)

case report form (CRF) or has an early discontinuation visit (EDV). A subject is classified as "completed" if this subject completes the full extent of the study as defined in the protocol at database lock.

A "discontinued" subject can be potentially slotted into the 3 periods of the study. The following algorithms will be used to slot the subject appropriately into the Evaluation Period, Down-Titration Period, and Post-Treatment Period.

- For Evaluation Period, the start date is the date of first dose of BRV, and the following algorithm is used to determine the end date:
  - If the subject enters the Down-Titration Period, then the date of EDV is the end date:
  - If the subject does not enter the Down-Titration Period but meets 1 of the following criteria, the Evaluation Period ends on date of last dose of BRV,
    - Without an EDV but having a termination CRF,
    - With an EDV and having a termination CRF,
    - With an EDV and the date of EDV prior to the database lock date and having no termination CRF.
- A subject is considered entering Down-Titration Period only if the subject has an EDV and at least 1 dose of study drug after the date of EDV, the start date of Down-Titration Period is set as 1 day after the date of EDV, and the Down-Titration Period ends on date of last dose of BRV. A subject without an EDV but having a termination CRF or with an EDV but without any dosing of study drug after the EDV will not have the Down-Titration Period, and no artificial Down-Titration Period will be created for analysis.
- A subject is considered entering the Post-Treatment Period if the subject has at least 1 contact (scheduled visit, unscheduled visit, or telephone contact) after the date of last dose of BRV. The Post-Treatment Period starts 1 day after date of last dose of BRV irrespective of entering the Down-Titration Period, and there is no end date.

A "completed" subject can potentially have Evaluation Period, Down-Titration Period, and Post-Treatment Period. At the time of study termination by the Sponsor, subjects will discontinue the study drug following the down titration process or will be converted without titration to commercial BRV where available; alternatively, subjects may be initiated without down-titration in a managed access program, named patient program, compassionate use program, or similar type of access program as allowed per country specific requirements in addition to legal and regulatory guidelines.

#### Monthly time intervals 3.2.5

A month is defined as 30 days and time intervals based on monthly durations are defined as a g di date on application and any extension application multiple of 30 days (eg. 12 months is defined as 360 days). The following definitions of 3-month and 6-month intervals are based on 30-day months where the date of first dose of BRV is Day 1:

| <b>Duration Definiti</b> |
|--------------------------|
| Days 1-90 |
| Days 91-180 |
| Days 181-270 |
| Days 271-360 |
| Days 1-180 |
| Days 181-360 |
| Days 361-540 |
| Days 541-720 |

Subsequent 3- and 6-month intervals are defined in a similar manner.

Six-month intervals are defined for the evaluation of direct and indirect cost parameters. Statistical summaries for direct and indirect cost parameters will only present results through the first 2 years of treatment. Three-month intervals will be used for analysis of efficacy outcomes and AEs.

For the analysis of efficacy outcomes, a subject is included in the analysis for a 3-month interval if the end date is on or after the *last day* of the 3-month interval and the subject diary was completed for at least 1 day during the 3-month interval.

For the analysis of AEs, a subject is included in the analysis for a 3-month interval if the end date is on or after the first day of the 3-month interval.

# Last Value on BRV Treatment

Last Value for QOLIE-31-P, HADS, EQ-5D, and socio-professional data is the last assessment strictly after the date of first dose of BRV and up to and including the YEV at the end of the second year and any EDVs for subjects who did not complete through the YEV at the end of the second year.

Last Value for clinical laboratory parameters, vital signs, and ECGs is the last available result obtained after the first dose of BRV and prior to or on the date of last dose of BRV. All

scheduled and unscheduled assessments within this time period will be considered. Last Value will be determined separately for each laboratory parameter.

#### 3.2.7 **Exposure duration and exposure duration cohorts**

Its ations thereof. At the final analysis, the overall duration of exposure (or On Treatment Period) will be calculated as the date of last dose of BRV minus the date of first dose of BRV plus 1 day. Each subject will be classified into one or more of the following exposure duration cohorts based on the duration of BRV exposure as calculated above:

All subjects >1 day >3 months ≥90 days >6 months ≥180 days >12 months  $\geq$ 360 days

This categorization will continue in 6-month increments past 12 months up to a time point that will be determined based on cumulative exposure at the time of the database lock.

#### 3.2.8 Study visit cohorts

Study visit cohorts are defined for summaries of QOLIE-31-P, HADS, and EQ-5D. Sixmonth, 12-month, 18-month, and 24-month cohorts are defined. Subjects will be classified into a study visit cohort if they attend the scheduled visit at the time point defined by the cohort. For example, subjects will be included in the 18-month study visit cohort if they attend the scheduled visit at 18 months (ie, FEV at Month 18). Subjects may be classified in more than 1 cohort. Generally, subjects included in a cohort for a later visit will be included in all earlier study visit cohorts (eg. 6-month and 12-month study visit cohorts for subjects in the 18-month study visit cohort), although this may not be the case in the event of a missed visit or if an unscheduled visit is conducted in lieu of a scheduled visit.

### **Definition of Baseline Values** 3.3

Baseline for all study outcomes will be based on baseline from the previous studies. For assessments performed at scheduled and unscheduled visits, Baseline will generally be the last result obtained or prior to the randomization visit of the previous study. Baseline will be defined separately for each hematology, blood chemistry, and urinalysis parameter.

Baseline for the evaluation of seizure frequency and seizure days will be calculated from the core study seizure diary based on the rules defined in Section 3.8.1.

#### 3.4 **Protocol deviations**

The criteria for identifying important protocol deviations and the classification of important protocol deviations will be defined separately in the Specification of Protocol Deviations document. Whenever possible, criteria for identifying important protocol deviations will be implemented algorithmically to ensure consistency in the classification of important protocol deviations across all subjects.

### 3.5 Analysis Sets

### 3.5.1 Safety Analysis Set

The Safety Analysis Set will consist of all subjects who took at least 1 dose of study drug but not including subjects entering the study from N01315.

Summaries of demographics and baseline characteristics, medical history, AEDs, non-AEDs, HADS, study drug exposure, and safety outcomes will be provided for the Safety Analysis Set.

A Modified Safety Analysis Set will also be defined to consist of all subjects who took at least 1 dose of study drug including subjects entering the study from N01315. Demographic, ongoing medication and safety assessment listings will be provided based on the Modified Safety Analysis Set.

## 3.5.2 Efficacy Analysis Sets

Efficacy Analysis Sets will consist of all subjects who took at least 1 dose of study drug and have at least 1 seizure diary day during the Evaluation Period. Separate Efficacy Analysis Sets are defined for subjects with focal epilepsy from N01114, N01252, and N01254 and subjects with generalized epilepsy from N01254.

A subject will be excluded from the Efficacy Analysis Set for POS or PGS if either they did not receive at least 1 dose of BRV, or the clinical database indicates that the daily seizure diary was not completed for any days on or after the first dose of BRV and on or prior to the end date of the Evaluation Period (see Section 8).

Seizure outcomes will be summarized for either the Efficacy Analysis Set for POS or the Efficacy Analysis Set for PGS. Summaries of epilepsy history, QOLIE-31-P, and EQ-5D will be provided for the Efficacy Analysis Sets for both POS and PGS. No summaries of these outcomes will be provided for ULD subjects or subjects entering the study from N01315, but these data will only be provided in subject data listings.

## 3.6 Treatment Assignment and Treatment Groups

This is an uncontrolled study in which all subjects receive BRV in doses that are optimally adjusted for each subject. Generally, statistical summaries will present all subjects combined as a single treatment arm unless otherwise indicated.

# 3.7 Coding dictionaries

Medical history and AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). Medications will be coded using the World Health Organization Drug Reference List (WHO-DRL). Prior and concomitant medical procedures will not be coded.

#### 3.8 **Definitions of study-specific derived variables**

#### 3.8.1 Calculation of seizure frequency/days

#### 3.8.1.1 Initial seizure data processing

Each seizure code in the clinical database will be mapped to exactly 1 of the following codes based on the 1981 International League Against Epilepsy (ILAE) classification: I, IA, IA1, IA2, IA3, IA4, IB, IB1, IB2, IC, II, IIA, IIB, IIC, IID, IIE, IIF, or III.

With regard to cluster seizures, investigator sites are to report the number of cluster episodes rather than reporting the estimated number of individual seizures. Therefore, no imputation will be applied for the seizure counts corresponding to reports of cluster seizures.

#### Calculation of adjusted seizure frequency 3.8.1.2

The following derivations apply only to subjects with Partial Onset Seizures

Baseline POS frequency for seizure types I, IA, IB, IC, and for all seizure types (I+II+III) will be obtained from the Baseline Period of the previous double-blind study.

The total number of seizures for seizure types I, IA, IB, and IC, and the total number of seizures for all seizure types (I+II+III) will be calculated overall, by 3-month time intervals, and over the cohort interval for each exposure duration cohort. All seizure diary on or after the date of first dose of BRV and prior to or on the date of last dose of BRV will be considered for these calculations.

Twenty-eight day adjusted seizure frequency for seizure types I, IA, IB, and IC, and for all seizure types (I+II+III) will be calculated overall, within each 3-month time interval, and over each exposure duration cohort interval by dividing the total number of seizures for each seizure type by the number of days for which the diary was completed overall, within each 3-month interval, and within each exposure duration cohort interval, and multiplying the resulting value by 28.

### Calculation of adjusted seizure days 3.8.1.3

The following derivations apply only to subjects with Primary Generalized Seizures, based on the 1981 ILAE classification, Primary Generalized Seizures include the generalized seizure types and unclassified seizure types.

Baseline seizure days for seizure types II, IIA through IIF, and for all seizure types (I+II+III) will be obtained from the Baseline Period of the previous study.

The total number of seizure days for seizure types II, IIA through IIF, and the total number of Twenty-eight day adjusted seizure days for seizure tweet to seizure types (I+II+III) will be calculated overall, by 3-mon and the transfer of the cohort interval for each exposure duration cohort. The satisfactory data defined in the Section 3.8.1.2 for POS frequency will be considered.

Twenty-eight day adjusted seizure days for seizure types (I+II+III) seizure days for all seizure types (I+II+III) will be calculated overall, by 3-month time intervals, and over the cohort interval for each exposure duration cohort. The same seizure

Twenty-eight day adjusted seizure days for seizure types II, IIA through IIF, and for all seizure types (I+II+III) will be calculated overall, within each 3-month time interval, and over each exposure duration cohort interval by dividing the total number of seizure days for each seizure type by the number of days for which the diary was completed overall (ie, over the periods defined in the Section 3.8.1.2), within each 3-month interval, and within each exposure duration cohort interval, and multiplying the resulting value by 28.

The QOLIE-31-P is an adaptation of the original QOLIE-31 (Cramer et al, 1998). The QOLIE-31-P includes 30 items grouped into 7 multi-item subscales (seizure worry [5 items], overall quality of life [2 items], emotional well-being [5 items], energy/fatigue [4 items] and a health status item. The second continuous conti and a health status item. The QOLIE-31-P total score, subscale scores, and health status item score are calculated according to the scoring algorithm described below, with scores ranging from 0 to 100 and higher scores indicating better functioning. In addition to these 31 items, the OOLIE-31-P includes 7 items assessing the degree of "distress" associated with the topic of each subscale (ie, distress items) and 1 item asking about the relative importance of each subscale topic (ie, prioritization item).

### Subscale Scores

As a first step to calculating the subscale scores, the individual responses for the 30 subscale items are rescaled to a 0 to 100 scale with higher scores reflecting better functioning; the rescaled values for each item are defined in Section 13.1. Each subscale score is then calculated by summing the rescaled responses for that subscale and dividing by the number of items without a missing response. A subscale score will be calculated only if at least 50% of the items within the subscale are present.

### Total Score

Total score is calculated as a weighted sum of the subscale scores based on the weighting in Section 13.1. Total score will be missing if at least 1 subscale score is missing. Total score will range from 0 to 100 with a higher score reflecting better functioning.

### Health Status Item

Responses for the health status item is a multiple of 10 ranging from 0 to 100 with a higher score corresponding to a better health status. The health status item response is analyzed without rescaling.

# Distress Items

Each subscale includes 1 distress item. The response for each distress item is an integer ranging from 1 to 5. The response for each distress item will be converted to a 0 to 100 scale (ie, 0.25, 50, 75, and 100) with a higher score corresponding to greater distress.

### Prioritization Item

The response for each subscale for the prioritization item is an integer ranging from 1 to 7. The prioritization ranking is analyzed without rescaling.

### 3.8.3 HADS

The HADS assessment consists of 14 items that are each scored on a 4-point scale ranging from 0 to 3, with a higher score corresponding to worse anxiety or depression. The depression and anxiety scores will be calculated by summing the scores for the items corresponding to each subscale, as described in the Hospital Anxiety and Depression Scale Manual (Snaith and Zigmond, 1994): the depression score is calculated as the sum of all even-numbered items; the anxiety score is calculated as the sum of all odd-numbered items. Scores for each subscale range from 0 to 21, with higher scores corresponding to a greater level of anxiety or depression.

Missing items will be replaced by the mean of non-mixed.

Missing items will be replaced by the mean of non-missing items from the same subscale when calculating the above, provided at least 50% of the items (ie, at least 4 of 7 items) within the subscale are present. A subscale score will not be calculated if more than 50% of the items are missing within a subscale. This rule applies separately to the subscale scores for anxiety and depression; for example, it may be possible to calculate the depression score in cases where the anxiety score is not calculated due to non-response.

## 3.9 Subject site transfers

Subjects may have transferred from one site to another through the course of participation in the study. Subjects that transferred from one site to another site, for whatever reason, have generally retained their subject number. However, in some cases, the subject number changed. When this is true, the most recently assigned subject number will be used for analyses and subject data listings. A record of any change in subject numbers will be presented in the Section 13.2.

## 4 STATISTICAL/ANALYTICAL ISSUES

## 4.1 Adjustments for covariates

No statistical testing is planned, therefore, this section is not applicable.

## 4.2 Handling of dropouts or missing data

Seizure frequency (subjects with POS) and seizure days (subjects with PGS) will be calculated over non missing diary days during each study period or time interval as described in Section 3.2.4 and Section 3.2.5; diary days for which seizure data were not obtained will not be considered in the calculation of seizure frequency or seizure days. Because the evaluation of efficacy is not the primary objective of this study, and because this is an uncontrolled study in a variable setting, which allows individualized optimization of dosing of BRV and concomitant AEDs, no summaries assessing the impact of missing seizure diary days are planned.

For subjects who prematurely discontinue during the Evaluation Period, the calculation of POS frequency and PGS seizure days will be based on available seizure diary while the subject was receiving BRV. The presence of such dropouts may influence the evaluation of the long-term outcomes for subjects who either do not discontinue or do not discontinue early in the study. Therefore, as described below, selected summaries will be produced by exposure

Brivaracetam

duration cohorts to allow an assessment of long-term outcomes without the potentially confounding influence of earlier discontinuations.

### 4.3 Interim analyses and data monitoring

Interim summaries were produced to support regulatory submissions for marketing authorization while this study is ongoing. There are no statistical concerns with such interim assessments for this study design.

#### 4.4 **Multicenter studies**

Efficacy and safety outcomes will not be assessed for individual investigator sites due to the No statistical testing is planned; therefore, this section is not applicable.

4.6 Use of an "Efficacy Subset" of subjects who are

All subjects who receive at least 1 dose of study drug and have at least 1 seizure diary day during the Evaluation Period will be included in efficacy summaries. Separate Efficacy Analysis Sets are defined for subjects with focal epilepsy from N01114, N01252, and N01254 and subjects with generalized epilepsy from N01254.

### Active-control studies intended to show equivalence 4.7

This section is not applicable for this study.

### 4.8 **Examination of subgroups**

Selected summaries will be provided for the following subgroups as specified within each of the following sections:

Two mappings of countries to regions are defined, 1 based on the classification requested by Food and Drug Administration (FDA), and 1 based on the regional classification for the CHMP (Committee for Medicinal Products for Human Use).

Countries will be mapped to geographic regions as follows for the FDA:

| Geographic Region (FDA) | Country |
|---|---|
| North America | Canada, United States, Puerto Rico |
| Latin America | Brazil, Mexico |
| Western Europe | Austria, Belgium, Finland, France, Germany, Ireland, |
| acili | Italy, Netherlands, Norway, Réunion, Spain, Sweden, |
| | United Kingdom, Switzerland |
| Eastern Europe | Bulgaria, Czech Republic, Estonia, Latvia, Hungary, |
| | Lithuania, Poland, Romania, Russia, Serbia and |
| | Montenegro, Turkey, Ukraine |
| Asia/Pacific/Other | Australia, Hong Kong, India, Israel, Japan, Singapore, |
| | South Africa, Republic of Korea, Taiwan, Tunisia |

Countries will be mapped to geographic regions as follows for the CHMP:

| Geographic Region | |
|---|---|
| (CHMP) | Country |
| North America | Canada, United States, Puerto Rico |
| Latin America | Brazil, Mexico |
| Europe (European Union | Austria, Belgium, Bulgaria, Czech Republic, Estonia, |
| [EU] member states) * | Finland, France, Germany, Hungary, Ireland, Italy, |
| | Latvia, Lithuania, Netherlands, Norway, Poland, |
| | Réunion, Romania, Spain, Sweden, United Kingdom |
| Europe (non-EU member | Russia, Serbia and Montenegro, Switzerland, Furkey, |
| states) | Ukraine |
| Asia/Pacific/Other | Australia, Hong Kong, India, Israel, Japan, Singapore, |
| | South Africa, Republic of Korea, Taiwan, Tunisia |

<sup>\*</sup> EU member states plus Norway.

- Indication (Partial Onset Seizures, Primary Generalized Seizures, ULD)
- Randomized treatment in the previous study (placebo [PBQ], BRV)

# 5 STUDY POPULATION CHARACTERISTICS

## 5.1 Subject disposition

Due to differences in data format across studies, in order to facilitate summary of subject disposition, the reasons for discontinuation for individual studies will be collapsed as follows for summaries:

| I TELL C | CDE D |
|---|---|
| LTFU Category | CRF Reason |
| ADVERSE EVENT | ADVERSE EVENT |
| LACK OF EFFICACY | LACK OF EFFICACY |
| | LOSS OF EFFICACY |
| LOST TO FOLLOW-UP | LOST TO FOLLOW-UP |
| SUBJECT CHOICE | CONSENT WITHDRAWN |
| SUP | WITHDRAWAL OF CONSENT FOR PERSONAL |
| 2.0 | REASONS NOT RELATED TO AES |
| be used to s | WITHDRAWAL OF CONSENT FOR PERSONAL |
| | REASONS NOT RELATED TO AES OR LACK OF |
| * 10° | EFFICACY |
| OTHER | PROTOCOL VIOLATION |
| Car | OTHER REASON |
| | OTHER |
| MISSING | If subject discontinued the study and the termination CRF is |
| | not available |

Only 1 primary reason for discontinuation should have been reported. In the event that more than 1 reason is specified in the clinical database, both reasons will be summarized and a

footnote will be added to the summary table to indicate that at least 1 subject is counted for multiple reasons for discontinuation.

ns or variations thereof An overall summary of disposition will be provided for all enrolled subjects (ie, all subjects who signed informed consent). The following will be summarized:

- The number of subjects in the Safety Analysis Set
- The number of subjects excluded from the Safety Analysis Set
- The number of subjects completed the study
- The number of subjects discontinued from the study, including the reason for discontinuation. If subject discontinued the study and the termination CRF is not available, the reason for discontinuation will be reported as "MISSING".

Additionally, an overall summary of disposition will present the following for subjects in the Safety Analysis Set:

- The number of subjects completed the study
- The overall number of subjects discontinued and the number of subjects discontinued by primary reason for discontinuation. If subject discontinued the study and the termination CRF is not available, the reason for discontinuation will be reported as "MISSING".

Overall subject disposition will also be summarized by geographic region and indication for the Safety Analysis Set.

The number of subjects within each geographic region and the number of subjects with each indication will be summarized for the Safety Analysis Set.

Kaplan-Meier estimates of the percentage of subjects completing 3, 6, 12, 24, 36, 48, and 60 months of treatment with BRV will be provided. This analysis will be based on the duration of exposure to BRV as defined in Section 3.2.7. Subjects who have permanently discontinued will be analyzed as events on the last day of treatment with study drug; subjects who complete the study will be censored on the last day of treatment with study drug.

The date of first subject in (date of earliest Visit 1), date of last subject out (date of last scheduled or unscheduled visit), number of enrolled subjects, and the number of subjects in each analysis set or indication will be summarized overall and by investigator site. Subjects who transferred sites will be summarized according to their original site.

Overall summary of disposition will be provided for safety analysis set, in addition, a separate overall summary will also be provided for modified safety analysis set.

### **5.2** 6 **Protocol Deviations**

The number and percentage of subjects with at least 1 important protocol deviation will be summarized overall and by category of protocol deviation for the Safety Analysis Set.

### **DEMOGRAPHICS AND OTHER BASELINE** 6 CHARACTERISTICS

Demographics

Demographics summaries will be based on demographic data from follow-up studies for subjects who enrolled in a follow-up study that collected demographic data. Otherwise demographics summaries will be based on demographic data collected.

Age, age category (1)

group (see below), body weight (kg), height (cm), body mass index (BMI) (kg/m²), and BMI category (<18.5, 18.5 to <25, 25 to <30, 30 to <40,  $\ge40$ ) will be summarized for the Safety Analysis Set. Demographic data will be summarized overall and by subgroup for indication and geographic region.

Racial group was not collected in a consistent manner across studies. For this reason, racial group will be collapsed as follows for statistical summaries:

**CRF Racial Group** Category

American Indian/Alaskan Native American Indian/Alaskan

Native

Asian, Asian/Pacific Islander, Indian/Pakistani Asian

Black, African-American Black

Native Hawaiian or Other Pacific Islander Native Hawaiian or Other

Pacific Islander

White, Caucasian, Hispanic White Other, Other/Mixed, Mixed Race Other/Mixed

moreover, the overall racial group will be collapsed as follows for statistical summaries:

Category **Racial Group from Previous Study** 

White, Caucasian, Hispanic White Black, African-American Black

Asian, Native Hawaiian or Other Pacific Islander, Asian/Pacific Islander, Asian

Indian/Pakistani

Other American Indian/Alaskan Native, Other, Other/Mixed

All subjects should be classified into one of the above categories.

Racial group, ethnicity (Hispanic or Latino, Not Hispanic or Latino), and racial subgroup (Indian/Pakistani, Japanese, Other) were not collected in a consistent manner across all studies; these variables will be provided in subject data listings if available in the clinical data from the previous study but will not be summarized.

#### 6.2 Medical and procedure history

#### 6.2.1 **Medical history diseases**

resolved and ongoing conditions at the time of entry into the previous studies, will be summarized overall and by primary MedDRA system organ class (SOC) and preferred term (PT) for the Safety Analysis Set.

6.2.2 Procedure history and concomitant procedures are not as 1

#### 6.3 History of epilepsy

All of the following are summarized using data collected at the time of entry into the previous studies or from the Baseline Period of the previous studies.

#### 6.3.1 Etiology of epilepsy

The number and percentage of subjects with each type of etiology as specified on the CRF (genetic, congenital, etc) from the previous studies will be summarized for the Efficacy Analysis Sets for POS and PGS. A subject will be counted as having a particular etiology if that etiology was either confirmed or suspected based on the investigator's assessment.

### Epileptic seizure profile 6.3.2

The number and percentage of subjects experiencing each seizure type at any time prior to study entry will be summarized for the Efficacy Analysis Sets for POS and PGS. The following seizure types will be summarized: I, IA, IA1 through IA4, IB, IB1, IB2, IC, II, IIA through IIF, III. A subject with a history of a more specific seizure type will be counted in all higher levels of seizure types (eg., a subject with a history of IB1 seizures will be counted for seizure types I, IB, and IB1).

#### 6.3.3 Classification of epileptic syndrome

The number and percentage of subjects with each epileptic syndrome will be summarized for the Efficacy Analysis Sets for POS and PGS. This summary will include the number and percentage of subjects within the following categories: localization-related epilepsy; idiopathic, symptomatic, and cryptogenic localization-related epilepsy; generalized epilepsy; and idiopathic, symptomatic, and cryptogenic generalized epilepsy.

### 6,3,4 **Focus localization**

The number and percentage of subjects with each category of focus localization (unknown, frontal, temporal, parietal, occipital) will be summarized for the Efficacy Analysis Set for POS. Subjects may be counted in more than 1 category of focus localization. A category for no available data will be included in the summary to account for subjects from N01114 since focus localization was not obtained for subjects from N01114. Percentages will still be out of the full POS Efficacy Analysis Set, including subjects from N01114.

#### 6.3.5 History of epileptic seizures

or status epilepticus and quantitative summaries of epilepsy duration, age at onset of first seizure, and percent of life with epilepsy, will be summarized for the Efficacy Analysis Sets for POS and PGS.

6.3.6 Seizure types experienced during baseline of the The number and percent.

The number and percentage of subjects experiencing each seizure type during the Baseline Period will be summarized for the Efficacy Analysis Sets for POS and PGS based on the Baseline seizure diary data from the previous studies. The following seizure types will be summarized: I, IA, IB, IC, II, and IIA through IIF.

Subjects will be counted for all higher levels of seizure type categories corresponding to the seizure types or seizure sub-types reported on the CRF.

#### 6.4 Medications

Medications recorded on the Concomitant Medications CRF and the Concomitant Medications (AEDs only) CRF will be classified as either AEDs or non-AEDs based on the preferred drug name search criteria, which are documented outside of the SAP.

- The medication is not an AED if it does not meet the search criteria based on preferred drug name, regardless of which CRF is used for reporting the medication. However, further review will be performed for medications that are recorded on the Concomitant Medications (AEDs only) CRF but are not included in the AEDs search criteria;
- For non-benzodiazepine medications, if the medication meets the search criteria for an AED based on preferred drug name, then the medication will be classified as an AED regardless of indication and regardless of which CRF the medication is recorded on;
- For benzodiazepines (identified using the search criteria), if the benzodiazepine is recorded on the Concomitant Medications (AEDs only) CRF, then the benzodiazepine will be classified as an AED;
- For benzodiazepines (identified using the search criteria), if the benzodiazepine is recorded on the Concomitant Medications CRFs, then the benzodiazepine will not be classified as an AED.

After medications are classified as AEDs or non-AEDs, the standard date imputation algorithms for start and stop date of the medication and first dose and last dose of BRV in the study will be applied. If an AED was taken at any time during dosing with BRV, then the AED is classified as a concomitant AED.

#### 6.4.1 Non-AEDs taken at study entry

The number and percentage of subjects taking non-AED medications at study entry for the Number of previous AEDs

The number and percentage of subjects taking an AED prior to entry into the previous study will be summarized by WHO-DRL preferred drug name for the POS and PGS Efficacy Analysis Sets based on the following categorization: 0-1 AEDs 2.4 AEE

6.4.3 History of previous AEDs previous double-blind study will be summarized by WHO-DRL primary therapeutic group

The number and percentage of subjects who had taken at least 1 AED prior to entry into the previous study will be summarized overall and by WHO-DRL preferred drug name for the POS and PGS Efficacy Analysis Sets.

#### 6.4.4 AEDs taken at study entry

The number and percentage of subjects taking AEDs at study entry for the previous doubleblind study will be summarized by WHO-DRL preferred drug name for the POS and PGS Efficacy Analysis Sets.

#### **Concomitant AEDs** 6.4.5

A concomitant AED is an AED which was taken during administration of BRV, regardless of the start and stop date of the AED. The number and percentage of subjects taking concomitant AEDs will be summarized by WHO-DRL preferred drug name for the POS and PGS Efficacy Analysis Sets.

### **MEASUREMENTS OF TREATMENT COMPLIANCE** 7

Study drug compliance will not be assessed due to the complexities associated with the calculation and interpretation of study drug compliance for this study. Study drug dosing will be provided in subject data listings.

## **EFFICACY ANALYSES**

In general, all study outcomes based on seizure frequency will be summarized for the Efficacy Analysis Set for POS and all study outcomes based on seizure days will be summarized for the Efficacy Analysis Set for PGS. No efficacy summaries are provided for

described in detail in Section 3.8.1.2 and Section 3.8.1.3, respectively.

All summaries of efficacy data are descriptive: no state. The derivations of 28-day adjusted seizure frequency and 28-day adjusted seizure days are

All summaries of efficacy data are descriptive; no statistical testing will be performed.

## Statistical analyses of secondary efficacy variables

The following variables are summarized for the Efficacy Analysis Set for POS.

#### 8.1.1 Partial onset seizure frequency

Twenty-eight day adjusted POS frequency will be summarized with quantitative descriptive will include all subjects in the POS Efficacy Analysis Set. Similar summaries will be provided for the full cohort interval and by 3-month time intervals for each exposure duration cohort.

8.1.2 Percent reduction in POS frequency

Percent reduction in POS frequency from Baseline to the On Treatment Period will be calculated as follows, where On Treatment Period Frequency is the 28-day adjusted POS frequency during On Treatment Period and Reseline P statistics for all subjects for the Baseline Period, the On Treatment Period, and by 3-month

POS frequency during the Baseline Period of the previous study.

% Reduction = 
$$100 \times \frac{\text{Baseline Period Frequency} - \text{On Treatment Period Frequency}}{\text{Baseline Period Frequency}}$$

A similar calculation applies to each 3-month time interval over the On Treatment Period and for the cohort interval for each exposure duration cohort.

Percent reduction from Baseline for POS frequency will be summarized with quantitative descriptive statistics for the On Treatment Period, and by 3-month time intervals over the On Treatment Period. The summary over the On Treatment Period will include all subjects in the POS Efficacy Analysis Set. Similar summaries will be provided for the full cohort interval and by 3-month time intervals for each exposure duration cohort. Percent reduction from Baseline for POS frequency will be summarized in the same manner by geographic region.

### Responder outcome for POS frequency 8.1.3

Responders over the On Treatment Period are defined as subjects with a 50% or greater reduction in 28-day adjusted POS frequency from Baseline to the On Treatment Period. A similar calculation applies to each 3-month time interval over the On Treatment Period and for the cohort interval for each exposure duration cohort.

The number and percentage of responders for POS frequency will be summarized for the On Treatment Period, and by 3-month time intervals over the On Treatment Period. The summary over the On Treatment Period will include all subjects in the POS Efficacy Analysis Set. Similar summaries will be provided over the full cohort interval and by 3-month time intervals for each exposure duration cohort. Responder rates for POS frequency will be summarized in the same manner by geographic region.

# 8.2 Analysis of other efficacy variables his docume.2.1

### Subjects with partial onset seizures

All of the following variables are summarized for the Efficacy Analysis Set for POS.

### 8.2.1.1 Specified Month seizure freedom

The numbers and percentages of subjects who are seizure free for all seizure types for any continuous 6-month interval, 12-month interval, 18-month interval, and so forth will be summarized overall for the period of time that subjects are being treated with BRV and by Exposure Duration Cohort. The overall summary will present the number and percentage of subjects who reported no seizures for the specified duration of seizure freedom and the seizure diary was completed for at least 90% of days within the seizure-free interval. Subjects whose duration of BRV treatment was less than the specified duration of seizure freedom will be considered failures for seizure-freedom. Summaries by exposure duration cohort will present the number and percentage of subjects who reported no seizures for the specified duration of seizure freedom at any time during the cohort interval (eg, through the end of Month 6 for the 6-month cohort) and the seizure diary was completed for at least 90% of days within the seizure-free interval. Percentages are relative to the number of subjects within each Exposure Duration Cohort.

A subject is seizure free for a 6-month interval if the subject did not report any seizures in the 6-month interval and the seizure diary was completed for at least 90% of days within the seizure-free interval. The percentage of days for which seizure diary was completed within a given 6-month interval will be calculated as follows based on a 30-day month:

% of days diary was done = 
$$100 \times \left[ \frac{180 - \text{number of days diary was not done in the interval}}{180} \right]$$

A similar calculation applies for 12-month seizure freedom based on 360 days, 18-month seizure freedom based on 540 days, and so forth.

### 8.2.2 Subjects with Primary Generalized Seizures

The following variables are summarized for the Efficacy Analysis Set for PGS.

### 8.2.2.1 All type seizure days

Twenty-eight day adjusted all other type seizure days will be summarized with quantitative descriptive statistics in the same manner as 28-day adjusted POS frequency.

## 8.2.2.2 Percent reduction in all type seizure days

Percent reduction in all other type seizure days from Baseline will be calculated in the same manner as percent reduction in POS frequency as described in Section 8.1.2. This variable will be summarized in the same manner as percent reduction in POS frequency.

## 8.2.2.3 Responder outcome for all type seizure days

Responder outcome for all other type seizure days will be derived in a manner similar to the responder outcome for POS frequency as described in Section 8.1.3. This variable will be summarized in the same manner as 50% responder outcome for POS frequency.

## 8.2.2.4 Specified month seizure freedom

Specified month seizure freedom for subjects in the PGS Efficacy Analysis Set will be derived in a manner similar to specified month seizure freedom for the POS Efficacy

Analysis Set as described in Section 8.2.1.1. This variable will be summarized in the same manner as specified month seizure freedom for subjects in the POS Efficacy Analysis Set.

#### 8.2.3 QOLIE-31-P

be provided for subjects with ULD. QOLIE-31-P was to be assessed at Months 2, 6, 12, 18, and 24 during the first 2 years of the Evaluation Period for subjects from N01252 and N01254, and assessments at Months 3, 6, 12, 18, and 24 during the first 2 years of the Evaluation Period for subjects from N01252 and N01254, and assessments at Months 3, 6, 12, 18, and 24 during the first 2 years of the Evaluation Period for subjects from N01252 and N01254, and assessments at Months 3, 6, 12, 18, and 24 during the first 2 years of the Evaluation Period for subjects from N01252 and N01254. at EDVs. The limited number of assessments obtained at Month 3 for N01114 will not be summarized but will be provided in subject data listings. Prior to Protocol Amendment 25, QOLIE-31-P may have been assessed for more than 2 years after study entry for some subjects. These additional assessments will not be summarized but will be provided in subject data listings.

Observed values for QOLIE-31-P total score and subscale scores for Seizure Worry, Daily Activities/Social Function, Energy/Fatigue, Emotional Well-Being, Cognitive Function, Medication Effects, Overall Quality of Life, and Health Status will be summarized for Months 2, 6, 12, 18, and 24 and Last Value for the Efficacy Analysis Sets for POS and PGS. For each time point, summary statistics will be presented for the baseline scores for subjects with a change from baseline at the time point in addition to summaries of the observed values and changes from baseline at each time point. Only subjects with a non-missing change from baseline will be summarized at each time point.

The above scores will be also summarized for the 6-Month, 12-Month, 18-Month, and 24-Month Study Visit Cohorts, including summaries of the baseline scores for all subjects within each study visit cohort and summaries of observed values and changes from baseline for each time point for each study visit cohort.

Similar summaries will be provided for QOLIE-31-P distress items Seizure Worry, Daily Activities/Social Function, Energy/Fatigue, Emotional Well-Being, Cognitive Function, Medication Effects, Overall Quality of Life. Only subjects with a non-missing change from baseline will be summarized at that time point.

The rankings of prioritization items (Seizure Worry, Daily Activities/Social Function, Energy/Fatigue, Emotional Well-Being, Cognitive Function, Medication Effects, and Overall Quality of Life) will be summarized at the same time points as above and for all subjects and by study visit cohort as defined above. Changes from baseline will not be summarized, and only the numbers of subjects and sample means will be presented.

### 8.2.4 EQ-5D

EQ-5D (EuroQol Group, 2000) will be summarized for the POS and PGS Efficacy Analysis Sets. No summaries of EQ-5D will be provided for subjects with ULD. EQ-5D was to be assessed at Months 2, 6, 12, 18, and 24 during the first 2 years of the Evaluation Period for subjects from N01252 and N01254. Additionally, QOLIE-31-P was to be assessed at EDVs. EQ-5D was not routinely assessed for subjects from N01114. Prior to Protocol Amendment 25, EQ-5D may have been assessed for more than 2 years after study entry for some subjects. These additional assessments will not be summarized but will be provided in subject data

Efficacy Analysis Sets for POS and PGS. The number and percentage of subjects with each response will be summarized for each dimension and time point. Percentages will be relative to the number of subjects with a response to the dimension at that time point. Additionally, for each dimension and time point, the number and percentage of subjects with each response will be summarized for baseline for subjects with time point. Additionally, each dimension and time points. Month, and 24-Month Study Visit Cohorts, including summaries for baseline for all subjects within each cohort and summaries of observed responses for all time points for each cohort.

Observed values for the EQ-5D visual analog scale (VAS) score will be summarized for Months 2, 6, 12, 18, and 24 and Last Value for the Efficacy Analysis Sets for POS and PGS. For each time point, summary statistics will be presented for the baseline VAS score for subjects with a change from baseline at the time point in addition to summaries of the observed values and changes from baseline at each time point. Only subjects with a nonmissing change from baseline will be summarized at each time point.

EQ-5D VAS score will also summarized for the 6-Month, 12-Month, 18-Month, and 24-Month Study Visit Cohorts, including summaries of the baseline scores for all subjects within each study visit cohort and summaries of observed values and changes from baseline for each time point for each study visit cohort.

### Direct cost parameters 8.2.5

Direct costs data are collected based on concurrent medical procedures, healthcare provider consultations not foreseen by protocol, hospital stays, and ER visits. All direct cost parameters will be not summarized but will be provided in subject data listings.

#### Indirect cost parameters 8.2.6

### The number of school or working days lost will not be 8.2.7 summarized but will be provided in subject data listings. Socioprofessional data

Socio-professional data is collected at Month 12 and Month 24 and at EDVs. Prior to Protocol Amendment 25, socio-professional data may have been collected for more than some subjects. These additional subject data listings. Some subjects from N01114 and subjects with ULD.

9 PHARMACOKINETICS

Places 2 years after study entry for some subjects. These additional assessments will not be summarized but will be provided in subject data listings. Socio-professional data are not

### PHARMACOKINETICS AND PHARMACODYNAMICS

Plasma samples for BRV and concomitant AEDs and antimyoclonic drugs (AMDs) will no longer be obtained, as directed by the integrated protocol amendment 25. No summaries of

BRV or concomitant AED/AMD plasma levels will be provided; plasma levels will only be provided in subject data listings.

SAFETY ANALYSES

Safety is assessed with AEs, laboratory tests (blood chemistry, hematology, urinalysis, and pregnancy test), vital signs, body weight, ECGs, physical examination, neurological examination, mental status, and psychiatric status. Summary tables will 1 summary tables will 1 summary tables will be provided for pregnancy testing, physical examination, neurological examination, mental status, or psychiatric status.

All safety summaries will be based on the Safety Analysis Set.

For subjects entering from N01315, their ongoing AEs will be transferred into N01125, and their safety assessments will be provided in subject data listings only, no summaries will be COPY applicati presented.

### 11.1 **Extent of exposure**

A daily dose will be calculated for each study day from the day of first dose of BRV to the day of last dose of BRV for the purposes of calculating modal dose. Daily dose will be calculated as the sum of the AM and PM dose for each day.

Modal daily doses will be calculated across all study days on or after the day of first dose of BRV and up to and including the day of last dose of BRV. Modal daily dose is the most frequently taken daily dose during this period. In the event of a tie, the modal dose will be set to the lower of the tied doses. Modal daily dose will be categorized as follows:

| Category | Definition |
|------------|--------------------------------|
| 5 mg/day | <20mg/day |
| 20mg/day 🐶 | ≥20mg/day to <50mg/day |
| 50mg/day | ≥50mg/day to <100mg/day |
| 100mg/day | $\geq$ 100mg/day to <150mg/day |
| 150mg/day | ≥150mg/day to <200mg/day |
| 200mg/day | ≥200mg/day |

Subject years of exposure will be calculated by summing the exposure duration in days for all subjects being summarized, and dividing the resulting value by 365.25.

Subject years of exposure will be presented overall and by modal dose for the Safety Analysis Set. The subject years of exposure presented by modal dose will be the total subject years of exposure of subjects with that modal dose.

The number and percentage of subjects exposed to BRV will be summarized overall and by modal dose category. The number and percentage of subjects in each Exposure Duration Cohort ( $\geq 3$  months,  $\geq 6$  months,  $\geq 12$  months, and so forth) will be summarized.

The number and percentage of subjects within each modal dose category will be summarized for each Exposure Duration Cohorts; percentages will be relative to the total number of subjects in each Exposure Duration Cohort.

In addition to the overall summaries of the above, the above will also be summarized by subgroup for region (North America, Europe [EU member states], Europe [non-EU member states], Asia/Pacific/Other), and by indication (Partial Onset Seizures, Primary Generalized Seizures, ULD).

### 11.2 Adverse events

## 11.2.1 Definition of treatment-emergent AE

AEs will be classified as either pre-study or treatment-emergent. Pre-study AEs are defined as AEs which had onset prior to the date of the first dose of BRV. TEAEs are defined as AEs that had onset on or after the day of first BRV dose. AEs with an incomplete onset date will be classified as TEAEs if the month and year of onset (when only the month and year are specified) is the same as the month and year of the first BRV dose or the year of onset (when only year is specified) is the same as the year of first BRV dose.

## 11.2.2 General summaries of TEAEs,

Pre-treatment AEs will be provided in a subject data listing; no summaries of pre-treatment AEs are planned.

An overall summary of AEs will provide the overall number of TEAEs and the numbers and percentages of subjects with at least 1 TEAE, with a TEAE that led to permanent discontinuation of study drug, with a drug-related TEAE, with a severe TEAE, with a treatment-emergent SAE, and with a drug-related treatment-emergent SAE. The number and percentage of subjects who died will also be summarized. This summary will be provided for all subjects in the Safety Analysis Set and also by subgroup for geographic region and indication.

The following summaries of TEAEs will be provided by MedDRA SOC and PT. All summaries are for the combined Evaluation, Down-Titration, and Post-Treatment Periods unless otherwise indicated.

Overall Incidence Summaries

- Incidence of TEAEs
- Incidence of TEAEs by 3-month time interval
- Incidence of TEAEs by study period (Evaluation, Down-Titration, Post-Treatment)
- Incidence of TEAEs for TEAEs occurring in at least 5% of subjects

- Incidence of TEAEs by 3-month time intervals for TEAEs occurring in at least 5% of subjects overall

A subject is included in a 3-month interval if the subject was receiving BRV at any time during that interval based on their duration of exposure to BRV (eg, a subject with exposure for 91 days is included in the time interval for Months 1-3 and Month.

AEs by 3-month intervals will include all subject was receiving as defined above. TFAE Incidence of TEAEs by maximum intensity
Incidence of drug-related TEAEs

erious Adverse Events
Incidence of treatment-emergent SAEs

Discontinuations due to TEAE

Incidence of TEAEs leading to permanent discontinuation of study drug included in summaries by 3-month time intervals.

Maximum Intensity and Causality

Serious Adverse Events

Discontinuations due to TEAE

TEAEs of interest

AEs of interest will be identified based on MedDRA search criteria, which are documented outside of the SAP. The following summaries will be provided for AEs of interest:

- Incidence of TEAEs of interest
- Incidence of TEAEs of interest by 3-month time interval

For the summary by maximum intensity, each subject will be counted at most once per SOC or PT according to the maximum intensity of all AEs within that SOC or PT. Severe intensity will be assumed for AEs for which intensity is not specified.

Drug-related AEs are AEs for which the relationship to study drug is specified as Related or AEs for which relationship is not specified.

### 11.30 **Clinical laboratory evaluations**

Clinical laboratory parameters (blood chemistry, hematology, urinalysis) are assessed at all FEVs, YEVs, EDVs, and at FV, and may also be assessed at Unscheduled Visits.

For subjects entering the study from N01315, the clinical laboratory assessments will be provided in subject data listings only. The baseline assessment of these subjects will not be carried over from the previous studies.
## 11.3.1 Hematology and blood chemistry parameters

Observed values for each planned hematology and blood chemistry parameter will be summarized for Baseline, Study Entry, and each scheduled visit during the Evaluation Period for which laboratory parameters were assessed, Last Value, EDV, and FV. Change from Baseline will be summarized for all post-Baseline time points including EV. Only laboratory parameters planned per protocol will be summarized; results for laboratory parameters not planned per the protocol will only be provided in subject data listings.

The number and percentage of subjects with an on-treatment potentially clinically significant treatment-emergent (PCST) value, PCST low value, and PCST high value will be summarized. This summary will consider all assessments after the first dose of BRV and prior to or on the date of the last dose of BRV.

Additionally, the number and percentage of subjects with a PCST value, PCST low value, and PCST high value will be summarized for Baseline, Study Entry, each visit during the Evaluation Period for which laboratory parameters were scheduled to be assessed, EDV, Last Value, and FV. Percentages for each parameter and time point will be relative to the number of subjects with a value at that time point.

PCST criteria (Sections 13.3.1 and 13.3.2) are based on FDA Division of Neuropharmacologic Drug Products guidelines with some UCB-defined additions.

Creatinine clearance, when available from the central laboratory, will be provided in subject data listings only and will not be summarized.

# 11.3.2 Macroscopic urinalysis

Quantitative urinalysis parameters will be summarized in the same manner as hematology and blood chemistry parameters. Response categories are negative, 1+, 2+, and 3+ for the qualitative urinalysis parameters occult blood, leukocytes, glucose, protein, and ketones and negative and positive for nitrates. Outcome values for these parameters are mapped to the levels Negative, 1+, 2+, and 3+ as follows for purposes of summary tables and the determination of PCST:

# Negative "Negative", "NEGATIVE", or other outcomes that clearly reflect a negative finding 1+ "1+", "+", "Trace", "TRACE", or other outcomes that clearly reflect trace amount 2+ "2+" or "++" 3+ "3+", "+++", or other outcomes that clearly reflect the data above 3+ (eg, "4+", "5+" etc) or more than 4 plus signs (eg, "++++", "+++++"etc)

For qualitative urinalysis parameters (occult blood, leukocytes, glucose, protein, ketones, and nitrates), the number and percentage of subjects with each response category will be summarized for Baseline, Study Entry, each scheduled visit during the Evaluation Period for

which urinalysis parameters were scheduled to be assessed, Last Value, EDV, and FV. Percentages for each parameter will be relative to the number of subjects with a result at each time point.

For occult blood, leukocytes, glucose, protein, ketones, and nitrates, the number and percentage of subjects with an on-treatment PCST value, PCST low value, and PCST high value will be summarized. This summary will consider all assessments after the first dose of BRV and prior to or on the date of the last dose of BRV.

Additionally, for occult blood, leukocytes, glucose, protein, ketones, and nitrates, the number and percentage of subjects with a PCST value, PCST low value, and PCST high value will be summarized for Baseline, Study Entry, each visit during the Evaluation Period for which laboratory parameters were scheduled to be assessed, EDV, Last Value, and FV. Percentages for each parameter and time point will be relative to the number of subjects with a value at that time point.

# 11.3.3 Microscopic urinalysis

In microscopic urinalysis, a small sample of urine is centrifuged to remove the liquid. The sediment is then examined under a microscope. In the urinalysis laboratory test group, other than urinalysis parameters such as Bilirubin, Blood, Glucose, Ketone, Nitrite, pH, Protein, Specific Gravity, Total protein, Hemoglobin, Beta-HCG, Occult Blood, and Leukocytes, a listing of microscopic analysis parameters will be provided; no summaries of microscopic analysis findings are planned.

# 11.4 Vital signs, physical findings, and other observations related to safety

For subjects entering the study from N01315, the vital signs, physical findings, and other observations related to safety assessments will be provided in subject data listings only. The baseline assessment from the previous studies of these subjects will not be presented.

# 11.4.1 Vital signs.

Vital signs are assessed at all FEVs, MEVs, YEVs, EDVs, and at FV, and may also be assessed at Unscheduled Visits. Body weight is assessed at all FEVs, YEVs, EDVs, and at FV, and may also be assessed at Unscheduled Visits.

Observed values for SBP, DBP, pulse rate, and body weight will be summarized for Baseline, Study Entry, each visit during the Evaluation Period for which vital signs or body weight were assessed, EDV, Last Value, and FV. Changes from Baseline for SBP, DBP, pulse rate, and body weight will be summarized for all post-Baseline time points.

The number and percentage of subjects with an on-treatment PCST value, PCST low value, and PCST high value will be summarized for SBP, DBP, pulse rate, and body weight. This summary will consider all assessments after the first dose of BRV and prior to or on the date of the last dose of BRV.

Additionally, the number and percentage of subjects with a PCST value, PCST low value, and PCST high value will be summarized for the above parameters for Study Entry, each visit

during the Evaluation Period for which vital signs or body weight were scheduled to be assessed, Last Value, EDV, and FV. Percentages will be relative to the number of subjects with a value at each time point.

Electrocardiograms

ECGs are assessed at all YEVs, EDVs, and at FV, and may also be assessed at Unscheduled Visits.

The number and percentage of subjects with no abnormality significant finding, and a clinically size in summary will a summary will consider all assessments after the first dose of BRV and prior to or on the date of the last dose of BRV.

Additionally, the number and percentage of subjects with no abnormality, an abnormal but not clinically significant finding, and a clinically significant finding will be summarized for Baseline, Study Entry, each visit during the Evaluation Period for which an ECG is scheduled to be performed, Last Value, EDV, and FV. Percentages will be relative to the number of subjects with an ECG assessment at each time point. Subjects are counted at most once at each time point based on the worst observed outcome across all abnormalities reported at that time point.

A subject number listing will be provided that identifies subjects with a clinically significant finding after the first dose of BRV for each type of ECG abnormality.

### Physical examination 11.4.3

A listing of abnormal physical examination findings will be provided; no summaries of physical examination findings are planned.

### 11.4.4 **Neurological examination**

A listing of neurological examination findings will be provided; no summaries of neurological examination findings are planned.

### 11.4.5 Psychiatric and mental status

A listing of abnormal Psychiatric and Mental Status findings will be provided; no summaries of Psychiatric and Mental Status findings are planned.

### 11.4.6° **HADS**

The scoring algorithm for HADS is described in 3.8.3.

During the first 2 years, HADS was assessed at Month 2, Month 6, Month 12, Month 18, and Month 24 and at EDV for subjects who discontinued the study prior to the YEV at the end of the second year for all subjects, and was also assessed at Month 4 and Month 9 for some subjects from N01114. HADS was not assessed for subjects from N01187 and N01236. Prior to integrated protocol amendment 25, HADS was being assessed for time points beyond the

YEV at the end of the second year. These additional assessments will not be summarized but will be provided in subject data listings.

Visit conort will only include scheduled visits up to the time of cutoff for the study visit cohort. Change from Baseline will be summarized at each visit during the Evaluation Period.

For summaries of observed values at each time point, only subjects with a charge Baseline value at that time point will be summarized. Observed values for HADS depression and anxiety scores will be summarized for Baseline

summary of change from Baseline.

### 11.4.7 **Columbia-Suicide Severity Rating Scale**

With global amendment 25 to the protocol, the Columbia-Suicide Seventy Rating Scale (C-SSRS) was added as an assessment at all study visits. Specific rules are provided to the study sites with regard to the identification of AEs or SAEs based on the outcome of this assessment. Because clinical events of interest will be recorded as AEs or SAEs, no study variable is defined for this assessment and no analyses are planned for the C-SSRS within the context of this study. However, subject data listings of the data for the C-SSRS will be provided. Additional listings will be provided for the subset of subjects with suicidal ideation and the subset of subject with actual suicide attempts.

Suicide ideation includes a "yes" answer to any 1 of the 5 suicidal ideation questions:



Suicide attempt includes response of a "yes" answer to any 1 of the 3 suicide attempt questions:



entory.

Jy the

July the grant and the present of the proper and the property of the property

### 13 **APPENDICES**

### 13.1 **QOLIE-31-P total and subscale score calculations**

| | | | Resp | onse | | | | Final Score |
|---|---|---|---|---|---|---|---|---|
| Scale/Item Numbers | 1 | 2 | 3 | 4 | 5 | 6 | Subtotal | 0-100 point scal |
| Seizure Worry | | | | | | | | Tel. |
| 30. | 0 | 20 | 40 | 60 | 80 | 100 | -1 | S, |
| 31. | 0 | 33.3 | 66.7 | 100 | _ | _ | ally | |
| 32. | 0 | 50 | 100 | | | | 29.0 | |
| 33. | 0 | 33.3 | 66.7 | 100 | _ | _ | 2 | |
| 34. | 100 | 75 | 50 | 25 | 0 | — <u>ij</u> i | | |
| | | | | | 1 | TOTAL: | Subtotal | ÷ 5 = |
| Overall Quality of Lif | | | | | 0 | 264 | | |
| 1. | | | response | ک by 10 | ), ~( | | | |
| 36. | 100 | 75 | 50 | 25 | 13:00. | | | |
| | | | | 1/2011 | | TOTAL: | | ÷ 2 = |
| Emotional Well-Being | g | | OP | | | | | |
| 7. | 0 | 20 | 40 | <b>∞</b> 60 | 80 | 100 | | |
| 8. | 0 | 20 | 240 (C) | <del>گ</del> 60 | 80 | 100 | | |
| 9. | 100 | 80 | 60 | | | | | |
| 10. | 0 | 20 | 40 | 60 | 80 | 100 | | |
| 11. | 100 | 80 0 | 60 | 40 | 20 | 0 | | |
| | | 20<br>80<br>80<br>80<br>80<br>20 | | | | TOTAL: | | ÷ 5 = |
| Energy/Fatigue | 0 | | | | | | | |
| 2. | 100 | 80 | 60 | 40 | 20 | 0 | | |
| 3. | 100 | 80 | 60 | 40 | 20 | 0 | | |
| 4. | 0 | 20 | 40 | 60 | 80 | 100 | | |
| 5. | 0 | 20 | 40 | 60 | 80 | 100 | | |
| 4. 5. Cognitive Functioning | | | | | | TOTAL: | | ÷ 4 = |
| 0 18 | | | | | | | | |
| 19. | 0 | 20 | 40 | 60 | 80 | 100 | | |
| 20. | 0 | 33.3 | 66.7 | 100 | | | | |
| 21. | 0 | 20 | 40 | 60 | 80 | 100 | | |
| 22. | 0 | 20 | 40 | 60 | 80 | 100 | | |
| 23. | 0 | 20 | 40 | 60 | 80 | 100 | | |
| 24. | 100 | 75 | 50 | 25 | 0 | | | |
| | | | | | | TOTAL: | | ÷ 6 = |

| UCB<br>Statistical Analysis P | lan | | | Brivarac | etam | | 11 February 2019<br>N01125 |
|---|---|---|---|---|---|---|---|
| Medication Effects<br>28.<br>26.<br>27. | 0<br>100<br>100 | 33.3<br>75<br>75 | 66.7<br>50<br>50 | 100<br>25<br>25 | <br>0<br>0 | _<br>_ | <br><b>5</b> 4. |
| Daily Activities/So | | | | | | TOTAL : | <br>÷ 3 = |
| 13.<br>14.<br>15.<br>16.<br>17. | 0<br>0<br>0<br>100<br>100 | 20<br>25<br>25<br>75<br>75 | 40<br>50<br>50<br>50<br>50 | 60<br>75<br>75<br>25<br>25 | 80<br>100<br>100<br>0<br>0 | 100<br>—<br>—<br>—<br>— | ÷3= |
| | | | | | , | TOTAL : | <br>÷ 5 (\$) |

Total score is calculated as a weighted sum of the subscale scores based on the weighting shown below. Total score will be missing if at least 1 subscale score is missing. Total score will range from 0 to 100 with a higher score reflecting better functioning.

| | Final Scale | | |
|---|---|---|---|
| QOLIE-31-P Scale | | Weight | Subtotal |
| | Ry all | 0.00 | |
| Seizure worry (a) | × × | 0.08 = | |
| Overall quality of life (b) | × × | 0.14 = | |
| Emotional well-being (c) | × × | 0.15 = | |
| Energy/fatigue (d) | × × | 0.12 = | |
| Cognitive functioning (e) | × | 0.27 = | |
| Medication effects (f) | × | 0.03 = | |
| Daily activities/Social functioning (g) | × | 0.21 = | |
| Seizure worry (a) Overall quality of life (b) Emotional well-being (c) Energy/fatigue Cognitive functioning Medication effects Daily activities/Social functioning (g) TOTAL SCORE: Sum subtotals (a) through the state of the st | igii (g) | | |

# 13.2 Subject site transfers



19 May 2016 N01125 UCB Statistical Analysis Plan Brivaracetam

### 13.3 **PCST** criteria

13.3.1 Hematology parameters

| 13.3.1 | Hematology parameters | - Gle | |
|---|---|---|---|
| Parameter | UCB Conventional Units | SI Units | CF |
| Hematocrit | For 1 m to < 6 m: \( \le 25\% \) | For 1 m to $< 6$ m: $\le 0.25$ | 0.01 |
| | For 6 m to $< 2$ y: $\le 27\%$ | For 6 m to $< 2$ y: $\le 0.27$ | |
| | For 2 y to $< 4$ y: $\le 29\%$ | For 2 y to $< 4$ y: $\le 0.29$ | |
| | For 4 y to < 12 y: $\leq 32\%$ (Female[F]); $\leq 35\%$ (Male [M]) | For 4 y to $<$ 12 y: $\le 0.32$ (F); $\le 0.35$ (M) | |
| | For $\geq 12$ y: $\leq 32\%$ (F); $\leq 37\%$ (M) | For $\geq 12$ y: $\leq 0.32$ (F); $\leq 0.37$ (M) | |
| Hemoglobin | For $< 6 \text{ m}$ : $\leq 9.7 \text{ g/dL}$ | For < 6 m: ≤ 97 g/L | 10 |
| | For 6 m to $< 12$ y: $\le 10.0$ g/dL | For 6 m to $< 12$ y: $\le 100$ g/L | |
| | For $\geq 12$ y: $\leq 9.5 \text{ g/dL (F)}; \leq 11.5 \text{ g/dL (M)}$ | For $\geq 12$ y: $\leq 95 \text{ g/L (F)}; \leq 115 \text{ g/L (M)}$ | |
| Platelets | $\leq 75 \times 10^9 / \text{L or} \geq 700 \times 10^9 / \text{L}$ | $\leq$ 75 x 10 <sup>9</sup> /L or $\geq$ 700 x 10 <sup>9</sup> /L | Not applicable (N/A) |
| White Blood | For $< 17$ y: $\le 3.0 \times 10^9 / \text{L}$ or $\ge 20 \times 10^9 / \text{L}$ ; | For $< 17 \text{ y}$ : $\le 3.0 \times 10^9/\text{L or} \ge 20 \times 10^9/\text{L}$ ; | N/A |
| Cell (WBC) | For $\geq 17$ y: $\leq 2.8 \times 10^9 / \text{L or} \geq 16 \times 10^9 / \text{L}$ ; | For $\geq 17$ y: $\leq 2.8 \times 10^9 / \text{L}$ or $\geq 16 \times 10^9 / \text{L}$ ; | |
| Red Blood | | For $< 17$ y: $\le 2.5 \times 10^{12}/L$ | 1 |
| Cell (RBC) | For $< 17 \text{ y: } \le 2.5 \text{ x } 10^6/\text{mm}^3$<br>For $\ge 17 \text{ y: } \le 2.0 \text{ x } 10^6/\text{mm}^3 \text{ (F); } \le 2.5 \text{ x } 10^6/\text{mm}^3 \text{ (M)}$ | For $\geq 17$ y: $\leq 2.0 \times 10^{12}/L$ (F); $\leq 2.5 \times 10^{12}/L$ (M) | |
| Eosinophils | $\geq 10\% \text{ or } \geq 0.7 \times 10^9/L$ | $\geq 0.10 \text{ or } \geq 0.7 \text{ x } 10^9/\text{L}$ | 0.01 or N/A |
| Neutrophils | $\leq 15\% \text{ or } \leq 1.0 \text{ x } 10^9/\text{L}$ | $\leq 0.15 \text{ or } \leq 1.0 \text{ x } 10^9/\text{L}$ | 0.01 or N/A |
| Basophils | $\geq 5\% \text{ or } \geq 0.4 \times 10^9/L$ | $\geq 0.05 \text{ or } \geq 0.4 \text{ x } 10^9/\text{L}$ | 0.01 or N/A |
| Monocytes | $\geq 20\% \text{ or } \geq 1.5 \times 10^9/L$ | $\geq 0.20 \text{ or } \geq 1.5 \text{ x } 10^9/\text{L}$ | 0.01 or N/A |
| Lymphocytes | For 1 m to $< 6$ m: $\le 22\%$ or $\ge 80\%$ | For 1 m to $< 6$ m: $\le 0.22$ or $\ge 0.80$ | 0.01 |
| | $\leq 2.1 \times 10^9 / L \text{ or } \geq 8.5 \times 10^9 / L$ | $\leq 2.1 \times 10^9 / L \text{ or } \geq 8.5 \times 10^9 / L$ | N/A |
| | For 6 m to $< 2$ y: $\le 15\%$ or $\ge 80\%$ | For 6 m to $< 2$ y: $\le 0.15$ or $\ge 0.80$ | 0.01 |
| | $\leq 1.5 \times 10^{9} / L \text{ or } \geq 7.5 \times 10^{9} / L$ | $\leq 1.5 \times 10^9 / L \text{ or } \geq 7.5 \times 10^9 / L$ | N/A |
| | For 2 y to $< 12$ y: $\le 12\%$ or $\ge 80\%$ | For 2 y to $< 12$ y: $\le 0.12$ or $\ge 0.80$ | 0.01 |
| | $\leq 0.0 \text{ x } 10^9/\text{L or} \geq 7.5 \text{ x } 10^9/\text{L}$ | $\leq 1.0 \times 10^9 / L \text{ or } \geq 7.5 \times 10^9 / L$ | N/A |
| | For 12 y to $< 17$ y: $\le 10\%$ or $\ge 80\%$ | For 12 y to $< 17$ y: $\le 0.10$ or $\ge 0.80$ | 0.01 |
| | $\leq 0.5 \times 10^9 / \text{L or} \geq 5.5 \times 10^9 / \text{L}$ | $\leq 0.5 \times 10^9 / L \text{ or } \geq 5.5 \times 10^9 / L$ | N/A |
| | For $\ge 17$ y:<br>$\le 0.5 \times 10^9/L$ or $\ge 5.5 \times 10^9/L$<br>$\le 10\%$ or $\ge 80\%$<br>$\le 0.5 \times 10^9/L$ or $\ge 4.5 \times 10^9/L$ | For $\geq 17$ y: $\leq 0.10$ or $\geq 0.80$ | 0.01 |
| | $\leq 0.5 \times 10^9 / \text{L or} \geq 4.5 \times 10^9 / \text{L}$ | $\leq 0.5 \times 10^9 / L \text{ or } \geq 4.5 \times 10^9 / L$ | N/A |
| Confidential | Page <b>45</b> of <b>50</b> | | |
| | SUL | | |
| Confidential | III. | | |
| 20 <sup>C)</sup> | | | |
| :6 | | | |
| /// | | | |
| * | | | |

Page **45** of **50** 

UCB19 May 2016Statistical Analysis PlanBrivaracetamN01125

# 13.3.2 Blood chemistry parameters

| | 1 | | Ī | | 1 |
|---|---|---|---|---|---|
| Parameter | | UCB Conventional Units | | SI Units | CF |
| AST (SGOT) | $\geq$ 3 times of ULN | | $\geq$ 3 times of ULN | an's | N/A |
| ALT (SGPT) | $\geq$ 3 times of ULN | | $\geq$ 3 times of ULN | te | N/A |
| ALP | For < 17 y: | $\geq$ 2 times of ULN, if normal range | For < 17 y: | $\geq$ 2 times of ULN, if normal range | N/A |
| | | adjusted to the age range; | | adjusted to the age range; | |
| | For $\geq 17$ y: | $\geq$ 3 times of ULN | | $\geq$ 3 times of ULN | |
| GGT | $\geq$ 3 times of ULN, | if baseline value $\leq 3$ times of ULN | | , if baseline value $\leq 3$ times of ULN | N/A |
| BUN | ≥ 30 mg/dL | | ≥ 10.71 mmol/L | | 0.357 |
| Urea | ≥ 60 mg/dL | | ≥ 10.02 mmol/L | | 0.167 |
| Creatinine | For < 17 y: | $\geq$ 1.5 mg/dL; | For < 17 y: | $\geq$ 132.6 umol/L; | 88.4 |
| | For $\geq 17$ y: | $\geq$ 2.0 mg/dL | For ≥ 17 y: | ≥ 176.8 umol/L | |
| Creatinine | For < 12 y: | < 70 ml/min (Schwartz) <sup>(a)</sup> | For < 12 y: | < 70 ml/min (Schwartz) <sup>(a)</sup> | N/A |
| clearance (calc) | For ≥ 12 y: | | For ≥ 12 y: | < 70 ml/min (Cockroft) <sup>(b)</sup> | |
| Total<br>bilirubin | ≥ 2.0 mg/dL | < 70 ml/min (Cockroft) <sup>(b)</sup> | ≥ 34.2 umol/L | | 17.1 |
| Glucose | $\leq 50 \text{ mg/dL or} \geq 1$ | 80 mg/dL | ≤ 2.775 mmol/L or | $r \ge 9.99 \text{ mmol/L}$ | 0.0555 |
| Total Protein | | $\leq 3.6 \text{ g/dL or} \geq 7.8 \text{ g/dL}$ | For $\geq 1$ m to $< 6$ m | $1: \leq 36 \text{ g/L or} \geq 78 \text{ g/L}$ | 10 |
| | | y: $\leq 4.7 \text{ g/dL or } \geq 9.5 \text{ g/dL}$ | For $\geq 6$ m to $< 17$ | y: $\leq 47 \text{ g/L or} \geq 95 \text{ g/L}$ | |
| | For ≥ 17 y: | $\leq$ 4.5 g/dL or $\geq$ 9.0 g/dL | For ≥ 17 y: | $\leq 45 \text{ g/L or} \geq 90 \text{ g/L}$ | |
| Albumin | For < 17 y: | $\leq 2.4 \text{ g/dL or} \geq 6.5 \text{ g/dL}$ | For < 17 y: | $\leq$ 24 g/L or $\geq$ 65 g/L | 10 |
| | For $\geq 17$ y: | $\leq 2.5 \text{ g/dL or} \geq 6.5 \text{ g/dL}$ | For $\geq 17$ y: | $\leq 25 \text{ g/L or} \geq 65 \text{ g/L}$ | |
| Globulin | For < 17 y: | $\leq 1.2 \text{ g/dL or} \geq 5.0 \text{ g/dL}$ | For < 17 y: | $\leq 12 \text{ g/L or} \geq 50 \text{ g/L}$ | 10 |
| | For $\geq$ 17 y: | $\leq 1.5 \text{ g/dL or} \geq 5.0 \text{ g/dL}$ | For $\geq$ 17 y: | $\leq 15 \text{ g/L or} \geq 50 \text{ g/L}$ | |
| Sodium | For < 17 y: | $\leq 120 \text{ mEq/L or} \geq 155 \text{ mEq/L}$ | For < 17 y: | $\leq 120 \text{ mmol/L or} \geq 155 \text{ mmol/L}$ | 1 |
| | For $\geq$ 17 y: | $\leq$ 115 mEq/L or $\geq$ 155 mEq/L | For $\geq 17$ y: | $\leq 115 \text{ mmol/L or} \geq 155 \text{ mmol/L}$ | |
| Potassium | For < 17 y: | $\leq$ 3.0 mEq/L or $\geq$ 6.5 mEq/L | For < 17 y: | $\leq$ 3.0 mmol/L or $\geq$ 6.5 mmol/L | 1 |
| | For ≥ 17 y: | $\leq 3.0 \text{ mEq/L or} \geq 5.8 \text{ mEq/L}$ | For $\geq 17$ y: | $\leq 3.0 \text{ mmol/L or} \geq 5.8 \text{ mmol/L}$ | |
| Calcium | For < 17 y; | $\leq$ 7 mg/dL or $\geq$ 11.5 mg/dL | For < 17 y: | $\leq 1.75 \text{ mmol/L or} \geq 2.875 \text{ mmol/L}$ | 0.25 |
| | For $\geq 17$ y: | $\leq$ 7 mg/dL or $\geq$ 15.5 mg/dL | For $\geq 17$ y: | $\leq 1.75 \text{ mmol/L or} \geq 3.875 \text{ mmol/L}$ | |

Confidential


| UCB | | 19 May 2016 |
|---------------------------|--------------|-------------|
| Statistical Analysis Plan | Brivaracetam | N01125 |

| Uric Acid | For < 12 y: | ≥ 8 mg/dL | For < 12 y: | ≥ 475.84 umol/L | 59.48 |
|---|---|---|---|---|---|
| | For $\geq 12$ y: | $\geq$ 8 mg/dL (F); $\geq$ 9.5 mg/dL (M) | For $\geq$ 12 y: | $\geq$ 475.84 umol/L (F); $\geq$ 565.06 umol/L | |
| | | | (M) | | |
| Cholesterol | ≥ 300 mg/dL | | ≥ 7.77 mmol/L | 'KEN' | 0.0259 |
| HDL | $\leq$ 25 mg/dL | | $\leq 0.65 \text{ mmol/L}$ | et | 0.0259 |
| LDL | $\geq$ 200 mg/dL | | ≥ 5.18 mmol/L | Kna | 0.0259 |
| Triglycerides | ≥ 300 mg/dL | | ≥ 3.42 mmol/L | 8.0 | 0.0114 |

<sup>(</sup>a) Schwartz equation (patients <12): Cr Cl ml/min = [Height (cm) \* 0.55] / serum creatinine


<sup>(</sup>b) Cockroft equation (patients ≥12): Male: Cr Cl ml/min = [(140-age) x body weight (kg)] (72 x serum creatinine),

Female: Cr Cl ml/min =  $[(140\text{-age}) \times \text{body weight (kg)}] / (72 \times \text{serum creatinine})] \times 0.85$ 

ALT=alanine aminotransferase; ALP=Alkaline phosphatase; AST=aspartate aminotransferase; BUN=blood urea nitrogen; CR CL=creatinine clearance; GGT=Gamma-glutamyl transpeptidase; HDL=High-density lipoprotein; LDL=low-density lipoprotein; SGOT=serum glutamic oxaloacetic transaminase; SGPT=serum glutamic pyruvic transaminase; ULN=Upper Limit of Normal.

### 13.3.3 **Urinalysis**

results in a five-point scale into a four-point scale, the lowest two positive results will be combined (see example below). For results reported with a scale of more than five-point, please consult your study physician for how to collapse into four-point scale.

Original Five-point Scale

Negative/None
Trace/T Qualitative urine parameters are generally reported by a descriptive score, which differs poin and any extensions of bpr

Trace/Rare/Mild/A Few Trace/1+/Rare/Mild/A Few

2+/Mod2+/Mod3+/Sev 3+/Sev

### 13.3.4 Vital signs and body weight

| Pulse rate | For 1 m to < 12 m. $\le$ 110 bpm and a decrease of $\ge$ 20 bpm from baseline or $\ge$ 180 bpm and an increase of $\ge$ 20 bpm from |
|---|---|
| | baseline baseline |
| | For 12 m to $<$ 3 y: $\leq$ 90 bpm and a decrease of $\geq$ 20 bpm from |
| | baseline or $\geq 150$ bpm and an increase of $\geq 20$ bpm from baseline |
| × | For 3 y to < 12 y: $\leq$ 65 bpm and a decrease of $\geq$ 20 bpm from baseline or $\geq$ 130 bpm and an increase of $\geq$ 20 bpm from baseline |
| ot be used to support | For 12 y to < 17 y: $\leq$ 60 bpm and a decrease of $\geq$ 20 bpm from baseline or $\geq$ 120 bpm and an increase of $\geq$ 20 bpm from baseline |
| not be used | For $\geq$ 17 y: $\leq$ 50 bpm and a decrease of $\geq$ 30 bpm from baseline or $\geq$ 120 bpm and an increase of $\geq$ 30 bpm from baseline |

bpm=Beats per minute. This document

| Systolic blood pressure | For 1 m to < 12 m: < 60 mmHg and a decrease of > 20 mmHg from baseline or > 110 mmHg and an increase of > 30 mmHg from baseline |
|---|---|
| | For 12 m to < 6 y: < 70 mmHg and a decrease of > 20 mmHg from baseline or > 120 mmHg and an increase of > 30 mmHg from baseline |
| | For 6 y to < 13 y: < 70 mmHg and a decrease of > 20 mmHg from baseline or > 130 mmHg and an increase of > 30 mmHg from baseline |
| | For 13 y and < 17 y: < 90 mmHg and a decrease of > 20 mmHg from baseline or > 140 mmHg and an increase of > 30 mmHg from baseline |
| | For $\geq$ 17 y: < 90 mmHg and a decrease of $>$ 30 mmHg from baseline or $>$ 180 mmHg and an increase of $>$ 40 mmHg from baseline |
| Diastolic blood pressure | For 1 m to < 12 m: < 40 mmHg and a decrease of > 15 mmHg from baseline or > 60 mmHg and an increase of > 20 mmHg from baseline |
| | For 12 m to < 6 y: < 45 mmHg and a decrease of > 15 mmHg from baseline or > 80 mmHg and an increase of > 20 mmHg from baseline |
| | For 6 y to < 13 y: < 50 mmHg and a decrease of > 15 mmHg from baseline or > 85 mmHg and an increase of > 20 mmHg from baseline |
| , IROTE S | For 13 y to < 17 y: < 55 mmHg and a decrease of > 20 mmHg from baseline or > 90 mmHg and an increase of > 30 mmHg from baseline |
| Le lised to sur | For $\geq$ 17 y: $<$ 50 mmHg and a decrease of $>$ 20 mmHg from baseline or $>$ 105 mmHg and an increase of $>$ 30 mmHg from baseline |
| Weight | For < 17 y: < 3% or > 97% of the normal body weight growth curve ranges for the age at date of weight assessment <sup>(a)</sup> and gender; |
| "Web" | For $\geq 17$ y: change of $\geq 7\%$ of baseline weight |
| (a) Once the subject reaches 17 regardless of their age in the st | years of age use the body curve criteria of a 17-year old tudy. |
| <b>\'</b> | |

# 14 AMENDMENT(S) TO THE STATISTICAL ANALYSIS PLAN

19 May 2016

N01125

### Rational for the amendment

The primary purpose for the amendment is (1) include subjects entering the study from study N01315 into this statistical analysis plan; (2) remove rules and definitions based on data cutoffs for interim analyses; (3) remove the summary analysis for direct cost parameter and indirect cost parameters, and as well as Socio-professional data.

### Change #1 (global)

Removed all rules and definitions based on data cutoffs for interim analyses throughout SAP.

### Change #2 (global)

Added analysis plan for subjects entering the study from study N01315 throughout SAP.

### Change #3 (global)

Section 8.2.5 Direct cost parameters, Section 8.2.6 Indirect cost parameters, Section 8.2.7 Socio-professional data

Removed all direct/indirect cost parameters and socio-professional data summary analysis.

### Change #4

Section 2.4 Determination of Sample Size

Changed the sample size to include subjects entering from N01315.

### Change #5

Section 3.5.1 Safety Analysis Set

Modified Safety Analysis Set and added a modified Safety Analysis Set.

# Change #6

Section 13.2 Subject site transfers

Removed subjects

### Change #7

Removed signature page. Using e-signature approval process through Source Submission.


# **Approval Signatures**

| Name: | Approval N01125-SAP-Amendment-1 | |
|---|---|---|
| Version: | 1.0 | |
| <b>Document Number:</b> | CLIN-000130975 | idions |
| Title: | N01125-SAP-Amendment-1 | of Varie |
| Approved Date: | 25 Feb 2019 | cions |
| | | Approvals |
| | | A SINY O |
| | | of and |
| | | , dicatile |
| | Document | |
| Approval<br>Verdict: Approved | C. K. | Name: Capacity: Clinical Date of Signature: 11-Feb-2019 14:05:58 GMT+0000 |
| | OF DA STATE | Name: |
| Approval<br>Verdict: Approved | arke times | Capacity: Clinical<br>Date of Signature: 25-Feb-2019 20:26:08 GMT+0000 |
| *( | Support any marketing author | |
| used | | |
| 20° De | | |
| ox carri | | |
| O.I. | | |
| cume | | |
| scument cannot be used to | | |